The incidence of psychological comorbidities in paediatric and young adults with inflammatory bowel disease, and the impacts of mental health conditions on quality of life, disease severity and resource utilisation: a population-based cohort study in the UK

# Protocol

NCT number: NCT05206734

Study ID: P043

**Document Date:** 24th January, 2022

# **Project highlights**

- This study will provide the first UK-based population level analysis of the risk of psychological comorbidities in children, adolescents, and young adults with IBD. The data resulting from this project will provide a measure of the magnitude of any associations. These insights will be valuable for clinicians managing people IBD in this age range; allowing early interventions to be targeted to those most at risk, and potentially reducing the likelihood of more serious future mental health problems.
- The dataset available for use in this project is one of the highest quality primary care data sources available world-wide. It provides the complete coded primary care record with robust data on comorbidities and treatments. In the paediatric population complete records since birth are available for the majority of people.

Our in-house matching algorithm ensures a higher quality of case-control
matching than is available using any other existing statistical software or
tools. This is vital to produce reliable data and satisfy external peer review.
Matching within a population-based sample has additional advantages
over the use of secondary care cohorts, US claim-based datasets, or disease
registry datasets. These advantages include minimisation of bias in the
control group and the opportunity to select a comparator group affected by
another chronic condition.

# **Background**

Inflammatory bowel disease (IBD) comprises 3 main subtypes; ulcerative colitis (UC), Crohn's disease (CD) and IBD unclassified (IBDU). IBD develops at any age; with around 10% diagnosed in childhood.(1) Whilst UC is the most common subtype of IBD in adults, CD is more common in the paediatric IBD (PIBD) population. International trends have confirmed a global rise in the incidence of PIBD; in particular, a steep rise in the incidence of CD.(2) In Scotland, data shows a dramatic increase in PIBD, especially in incidence of CD which has risen 500% over just 40 years.(3)

PIBD is associated with more extensive disease compared to adult onset IBD, with additional considerations which include growth failure, delayed puberty, poor bone density and psychosocial impact during a vulnerable period of life.(1, 4) The goals of treating IBD are to induce and maintain remission and to avoid disease complications, drug-related complications and unnecessary surgery, psychological health, promoting a return to, and maintenance of, a normal lifestyle that includes education, family, social function and physical activity.(1, 5) Other essential goals in children include optimizing growth, puberty, and psychological health and promoting a return to, and maintenance of, a normal lifestyle that includes education, family, social function, and physical activity.(1)

Psychological comorbidities associated with PIBD include anxiety; which may be related to the perceived or actual side effects of IBD therapies, altered body image and a feeling of lack of control over their lives, and depression; associated with severe/active disease, current steroid use and the need for an ostomy.(6) Conflicting results and methodological constraints have limited previous understanding of psychosocial functioning in PIBD.(7) Reported rates of clinically significant symptoms of depression and anxiety have ranged from 25% to 73% in children and adolescents with PIBD.(6) However, recent studies highlight growing concerns for psychiatric morbidity in IBD in children and young adults. A US study(8) of 58,020 IBD patients aged 5-24 reported a prevalence of psychiatric disorders of 21.6%; mainly comprising depression and anxiety disorders. IBD was found to be 5 times more likely associated with psychiatric disorders than with controls, and the incidence of these disorders was associated with a steady increase in trend over time (2% in 2006 compared to 15% in 2017).(8) Similarly, Swedish data(9) from 6464 PIBD patients, indicate an association of IBD with psychiatric morbidity of 17.3%. Most concerningly, this study reported IBD to be significantly associated with suicide attempt and as well as mood disorders, disorders, disorders, eating personality disorders, deficit/hyperactivity disorder, and autism spectrum disorders. Results for each sex were similar. A correlation of age and development of psychiatric disorders was indicated for patients with very early-onset IBD (<6 years).

Furthering our understanding of the psychosocial sequalae of IBD in children and young adults is particularly important in light of evidence suggesting that symptoms of anxiety and depression may decrease adherence to treatment, thus impacting on longer term disease outcomes,(6) and has been emphasized in a recent call to action issued within gastroenterology to improve understanding and early identification of comorbidities associated with IBD.(10)

To the best of our knowledge, there have not been any large population-based studies assessing the association between psychosocial comorbidities in IBD in

children and young adults and disease related outcomes. The aim of this study is therefore to fill this data gap, and to examine the following objectives.

Such new insights will be valuable for clinicians in optimising patient care for IBD patients; allowing early interventions to be targeted to those most at risk, and potentially preventing the development of more serious mental health problems such as depression; linked to difficulties with medication adherence, and anxiety; which may exacerbate future disease activity.(7, 10)

Ultimately, we anticipate that these data will be useful in understanding the potential cycle and interrelationship between IBD and mental health in children and young adults.

### Objectives: Stream 1 - Incidence of mental health conditions

#### **Primary Objectives**

 Compare the risk and cumulative incidence of mental health conditions in children and young adults with IBD compared to matched population controls in the primary care setting, stratified by IBD type

#### **Secondary Objectives**

• Determine severity of mental health conditions in those with and without IBD (e.g. evidence of self-harm, suicide attempt, behavioural disorders)

# Objectives: Stream 2 - Impacts of mental health conditions

#### **Primary Objective:**

 Determine the association of mental health conditions in children and young adults with IBD on quality-of-life indicators

#### **Secondary Objectives:**

 Compare IBD severity/disease markers in children and young adults with IBD with and without mental health illness • Compare healthcare resource utilisation in children and young adults with IBD with and without mental health illness

## **Methods**

The study protocol was specified a priori and registered with ClinicalTrials.gov (Study identifier: NCT05206734).

#### Data source

The Optimum Patient Care Research Database (OPCRD). This database incorporates pseudonymised primary care records from 700 GP practices distributed across England, Wales, Scotland and Northern Ireland. The current OPCRD cohort size is over 5 million actively registered people, and historic records available for 10.1 million people. The cohort dataset can be enhanced through direct-to-patient and direct-to-care provider questionnaires at additional cost if required.

# Study design

The proposed study will use the retrospectively collected data of all eligible patients within the database at the date of data extraction. Within this primary care cohort, all patients with IBD comprising of the three main subtypes; ulcerative colitis (UC), Crohn's disease (CD) and IBD unclassified (IBDU), excluding microscopic colitis, radiation induced enterocolitis and drug-induced enterocolitis, will be identified using diagnostic codes and prescription records. A diagnostic algorithm will be developed to facilitate robust case identification of IBD and IBD subtypes, as well as mental health outcomes.

#### Statistical methods

We will use standard descriptive statistics (mean, standard deviations, etc) to describe the characteristics of the study cohort.

## Recorded sociodemographic characteristics and clinical features

Sociodemographic data will comprise by age group, age at diagnosis, gender, ethnicity, and socioeconomic status. Ethnicity will be categorised as follows to be consistent with the UK official census categories: White, Asian, Black African/Caribbean, Mixed, and Other. The index of multiple deprivation (IMD) will be used as a measure of socioeconomic status. This is derived from patient postcode at the point of data extraction.

## Stream 1: Study Cohort

#### Stream 1: Definition of people with new onset IBD

The eligible PIBD cases will comprise all incident cases of PIBD over the last decade, we will not follow patients up beyond 01/01/2020 due to changes in patient health behaviour and primary care interactions due to COVID-19. We will extract sociodemographic details for all these cases and matched controls (described below). Sociodemographic data will comprise by age group, gender, ethnicity, and socioeconomic status. Ethnicity will be categorised as follows to be consistent with the UK official census categories: White, Asian, Black African/Caribbean, Mixed, and Other. The index of multiple deprivation (IMD) will be used as a measure of socioeconomic status. This is derived from patient postcode at the point of data extraction.

#### Stream 1: Definition of matched controls without IBD

We will match each incident case of PIBD with controls (children without IBD) using propensity score matching (matching on the sociodemographic variables list above and matching within primary care practice if numbers allow). People with a known diagnosis of irritable bowel syndrome (IBS) will be excluded from the potential pool of controls. We will compare the incidence of new onset mental health conditions in PIBD and controls using a similar approach to that used by Butwick et al. (2019) in their paper exploring psychiatric disorders in a

PIBD cohort in Sweden.(9) The mental health conditions to be examined are listed in table 1 although there is scope to add to or modify these in discussion with the study authors. For a composite 'any psychological condition' outcome (see Table 1), risk will be stratified by age of PIBD onset and sex.

We will then go beyond the analysis of the Swedish study to estimate the cumulative risk of the 'any psychological condition' composite outcome in PIBD patients compared with controls. This will provide a unique, robust, estimate of the overall mental health burden (prevalence) in PIBD.

| Condition | Description |
|---|---|
| Primary outcomes | |
| Any psychological | A composite of all the chronic psychiatric conditions listed |
| condition | below* (depression, anxiety, eating disorders, body image |
| | disorder, attention-deficit disorder, behavioural disorders, |
| | adjustment disorder, acute stress disorder, and post-traumatic |
| | stress disorder) |
| Depression | Major recurrent depression or treated depressive episode |
| Anxiety | Non-phobia related anxiety episodes or disorder |
| Secondary outcomes | |
| Self-harm | Any coded episode of deliberate self-harm of any type |
| Suicide attempt | Any episode of suicide attempt and suicide related codes, |
| | including deliberate medication overdose |
| Other chronic psychiatric | Eating disorders, body image disorder, attention-deficit |
| conditions | disorder (ADHD), behavioural disorders, adjustment disorder, |
| | acute stress disorder, schizophrenia, bipolar disorder and post- |
| | traumatic stress disorder (PTSD) |
| Others | Problems with sleep |

<sup>\*</sup>this excludes conditions which are potentially single events i.e. self-harm or suicide attempt. (See Appendix 1 – Table s3 for Read Codes and SNOMED Codes

for mental health conditions, Table s4 for mental health condition algorithms and Table s5 for WHO ICD-10 mental health conditions).

#### Stream 1: Incidence of mental health conditions

The study will report the incidence of each mental health condition overall in the PIBD cases and controls, and adjusted hazard ratios to test the association between PIBD and risk of the same mental health conditions. Within the PIBD cohort we will examine the relationship between PIBD age of onset, sex, ethnicity, and social deprivation and the 'any psychological condition' composite outcome.

Cox proportional hazards models will be used to compare disease incidence in PIBD cases and controls and also when comparing the associations of baseline features and outcomes within the PIBD cohort. The study start date will be the date of diagnosis of PIBD or, for controls, the date of diagnosis of their matched counterpart. The end of follow-up will be the first of; the point of data extraction (exact date TBC), the patient's 25th birthday, date of loss to follow-up (either GP) practice deregistration or death). All individuals contributing at least six months of follow-up time in the analysis will be included. Those with existing evidence of the mental health condition prior to baseline will be excluded for analysis of that particular outcome where it would not reoccur, for example if individual has already received a diagnosis of recurrent depressive disorder they would not receive this diagnosis again, although conditions at baseline that can reoccur, such as suicide attempt, would not be excluded. Models will be adjusted for age, gender, socioeconomic status, ethnicity, and other childhood conditions (asthma, atopic dermatitis, allergic rhinitis, thyroid disease, epilepsy, diabetes, cancer, juvenile idiopathic arthritis (JIA) including systemic JIA, systemic lupus erythematosus (lupus), ankylosing spondylitis (AS) and psoriatic arthritis). Statistical significance for analyses will be reported using P values and 95% confidence intervals as appropriate.

Cumulative risk (i.e. prevalence) of the 'any psychological condition' composite outcome will be evaluated up to age 25. Cumulative incidence will be calculated by using methods to estimate risk similar to those recently published when assessing lifetime risk of other chronic conditions in the Lancet.(11, 12) Key outputs will be cumulative risk plots, presenting the cumulative incidence of the outcome by age for PIBD patients compared to controls. At a particular age, the cumulative incidence estimate can be interpreted as the lifetime incidence of the outcome up until the year of age in question. Childhood cumulative risk will be defined as the cumulative incidence at age 18.

### Stream 1: Sensitivity analysis

To evaluate the magnitude of potential bias from including, as matched controls, people who are registered with GP practices but who do not attend their practice, we also repeated the primary analysis including only controls with a least one primary care consultation in the year preceding their index date.

All statistical analyses were performed using R statistical package software version 3.4.1. The study was conducted in line with the RECORD (Reporting of studies conducted using observational routinely collected data) guidelines.(13)

#### Stream 2:

## Stream 2: Study design

The proposed study will use the retrospectively collected data of all eligible patients within the database at the date of data extraction. Within this primary care cohort, all patients with IBD will be identified using diagnostic codes and prescription records. A diagnostic algorithm will be developed to facilitate robust case identification of IBD and IBD subtypes as well as mental health outcomes.

## Stream 2: Study cohort

The eligible IBD cases will comprise all prevalent cases of IBD aged under 25 at 01/01/2015 (index date) comprising of the three main subtypes; ulcerative colitis (UC), Crohn's disease (CD) and IBD unclassified (IBDU), excluding microscopic colitis, radiation induced enterocolitis and drug-induced enterocolitis. We will extract sociodemographic details for all individuals. Sociodemographic data will comprise by age group, age at diagnosis, sex, ethnicity, and socioeconomic status. Ethnicity will be categorised as follows to be consistent with the UK official census categories: White, Asian, Black African/Caribbean, Mixed, and Other. The index of multiple deprivation (IMD) will be used as a measure of socioeconomic status. This is derived from patient postcode at the point of data extraction.

We will identify comorbid psychological condition groups in all people with PIBD. These will comprise 3 composite phenotypes; anxiety/panic disorders, major depression or depressive episodes, and other psychological conditions. Other psychological conditions will be a composite of; eating disorders, body image disorder, attention-deficit disorder (ADHD), behavioural disorders, adjustment disorder, acute stress disorder, schizophrenia, bipolar disorder and post-traumatic stress disorder (PTSD). Where numbers are sufficient, subgroups of the broad 'other psychological conditions' composite may be examined.

At the index date, we will define groups in the IBD case population based on mental health phenotype, including a comparator group without mental health comorbidity at the index date, and compare the sociodemographic characteristics of these groups.

## Stream 2: Follow-up

We will then describe incidence of each study outcome in the five years after the index date for each group, and the relative incidence of each outcome in those with and without mental health comorbidity.

## Stream 2: Study outcomes

These will comprise the following.

#### **Quality of life indicators:**

Affective symptoms (depression, low mood, deliberate self-harm, suicidal ideation or parasuicide), IBD symptoms, absence from school, absence from work, unemployment, substance abuse, and sleep problems. IBD symptoms will comprise; abdominal pain, discomforts or bloating, diarrhoea, weight loss, growth retardation and tiredness/fatigue. (See Appendix 1 – Table s1 for Read Codes and SNOMED codes).

#### **IBD** severity indicators:

Medication use, surgical intervention, nutritional supplement use, and markers of nutritional status. Surgical intervention will comprise any abdominal surgery, and stoma formation (as a separate outcome). Medication use will comprise use of: rectal 5-aminosalicylic acid (5-ASA), oral 5-ASA, rectal steroids, oral steroids, antimetabolites, tumour necrosis factor inhibitors (TNFi) and other biologic therapies. The latter of these groups may not be well captured in primary care and if so this will be reported in the limitations section of the final study manuscript. Nutritional supplements will comprise the five most prescribed nutritional supplements: Modulen, Fortisip, Ensure, Osmolite, and Neocate. Nutritional markers will comprise; being underweight (under the 5th centile of weight for height or BMI < 18.5 kg/m² after age 18) and growth retardation related codes. (See Appendix 1 – Table s2 for Read Codes and SNOMED codes).

#### Healthcare resource utilisation:

Primary care attendances and hospital admissions. Hospital admissions will be separated into general admissions (including those for IBD) and psychiatric admissions. (See Appendix 1 – Table s2 for Read Codes and SNOMED codes).

#### Stream 2: Statistical methods

We will use standard descriptive statistics (mean, standard deviations, etc) to describe the characteristics of the study cohort overall and by mental health phenotype. Across mental health condition phenotypes we will describe the incidence of recording of all the quality-of-life indicators, IBD severity markers, and healthcare resource utilisation outcomes up to five years after the index date (01/01/2015), compared to incidence in the group without mental health conditions. The end of follow-up will be the first of; 01/01/2020 (5 years after the index date) we will not follow patients up into 2020/21 due to changes in patient health behaviour and primary care interactions due to COVID-19, the patient's 25th birthday, date of loss to follow-up (either deregistration or death). All individuals contributing at least six months of follow-up time in the analysis will be included. We will not follow patients up into 2020/21 due to changes in patient health behaviour and primary care interactions due to COVID-19.

Relative incidence between those with and without mental health conditions will be estimated for repeated events (e.g. number of hospital admissions) and binary events (e.g. quality of life indicators) using, as appropriate, Poisson regression, negative binomial regression (if we need to account for overdispersion), or zero-inflated Poisson regression (if we need to model rare events). To account for variable duration of follow-up, we will include the natural logarithm of person-years of follow-up as a model offset. Confidence intervals will be estimated using robust SEs. Models will be adjusted for age, gender, socioeconomic status, ethnicity, and other childhood conditions (asthma, atopic dermatitis, allergic rhinitis, thyroid disease, epilepsy, diabetes, cancer, juvenile idiopathic arthritis (JIA) including systemic JIA, systemic lupus erythematosus (lupus), ankylosing spondylitis (AS) and psoriatic arthritis). Statistical significance for analyses will be reported using P values and 95% confidence intervals as appropriate.

Where numbers allow, we will report absolute and relative incidence in subgroups by, mental health condition group, age group (5-<12; 12-<16; 16-<18; 18-<25) (child, adolescent, young adult), and sex.

## References

- 1. Wilson DC, Russell RK. Overview of paediatric IBD. Seminars in Pediatric Surgery. 2017;26(6):344-8.
- 2. Benchimol EI, Fortinsky KJ, Gozdyra P, Van Den Heuvel M, Van Limbergen J, Griffiths AM. Epidemiology of pediatric inflammatory bowel disease: A systematic review of international trends. Inflammatory Bowel Diseases. 2011;17(1):423-39.
- 3. Henderson P, Hansen R, Cameron FL, Gerasimidis K, Rogers P, Bisset MW, et al. Rising incidence of pediatric inflammatory bowel disease in Scotland\*. Inflammatory Bowel Diseases. 2012;18(6):999-1005.
- 4. Grover Z, De Nardi A, Lewindon PJ. Inflammatory bowel disease in adolescents. Aust Fam Physician. 2017;46(8):565-71.
- 5. Turner D, Ricciuto A, Lewis A, D'Amico F, Dhaliwal J, Griffiths AM, et al. STRIDE-II: An Update on the Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE) Initiative of the International Organization for the Study of IBD (IOIBD): Determining Therapeutic Goals for Treat-to-Target strategies in IBD. Gastroenterology. 2021;160(5):1570-83.
- 6. Nasiri S, Kuenzig ME, Benchimol EI. Long-term outcomes of pediatric inflammatory bowel disease. Semin Pediatr Surg. 2017;26(6):398-404.
- 7. Ross SC, Strachan J, Russell RK, Wilson SL. Psychosocial functioning and health-related quality of life in paediatric inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2011;53(5):480-8.
- 8. Thavamani A, Umapathi KK, Khatana J, Gulati R. Burden of Psychiatric Disorders among Pediatric and Young Adults with Inflammatory Bowel Disease: A Population-Based Analysis. Pediatric Gastroenterology, Hepatology & Nutrition. 2019;22(6):527.
- 9. Butwicka A, Olén O, Larsson H, Halfvarson J, Almqvist C, Lichtenstein P, et al. Association of Childhood-Onset Inflammatory Bowel Disease With Risk of Psychiatric Disorders and Suicide Attempt. JAMA Pediatrics. 2019;173(10):969-78.
- 10. Argollo M, Gilardi D, Peyrin-Biroulet C, Chabot J-F, Peyrin-Biroulet L, Danese S. Comorbidities in inflammatory bowel disease: a call for action. The Lancet Gastroenterology & Hepatology. 2019;4(8):643-54.
- 11. Gershon AS, Warner L, Cascagnette P, Victor JC, To T. Lifetime risk of developing chronic obstructive pulmonary disease: a longitudinal population study. Lancet (London, England). 2011;378(9795):991-6.
- 12. Rapsomaniki E, Timmis A, George J, Pujades-Rodriguez M, Shah AD, Denaxas S, et al. Blood pressure and incidence of twelve cardiovascular diseases: lifetime risks, healthy life-years lost, and age-specific associations in 1·25 million people. Lancet (London, England). 2014;383(9932):1899-911.

13. Benchimol EI, Smeeth L, Guttmann A, Harron K, Moher D, Petersen I, et al. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. PLoS Med. 2015;12(10):e1001885.

# **Appendices**

# Appendix 1

**sTable 1.1.** Read and SNOMED codes to be used to identify cases of IBD and IBD subtypes

| Ulcerative Colitis (UC) | | |
|-------------------------|---------|------------------------------------------|
| Read V2 Code | Term ID | Description |
| J41 | All | Ulcerative colitis and/or proctitis |
| J410. | All | Ulcerative proctocolitis |
| J4100 | All | Ulcerative ileocolitis |
| J4101 | All | Ulcerative colitis |
| J4102 | All | Ulcerative rectosigmoiditis |
| J4103 | All | Ulcerative proctitis |
| J4104 | All | Exacerbation of ulcerative colitis |
| J410z | All | Ulcerative proctocolitis NOS |
| J411. | All | Ulcerative (chronic) enterocolitis |
| J412. | All | Ulcerative (chronic) ileocolitis |
| J413. | All | Ulcerative pancolitis |
| N0454 | All | Juvenile arthritis in ulcerative colitis |
| N0310 | All | Arthropathy in ulcerative colitis |
| Read CTV3 Code | Term ID | Description |
| XE0ag | All | Ulcerative colitis |
| XaZ2j | All | Left sided ulcerative colitis |
| XaYzX | All | Ulcerative pancolitis |

| XaK6E | All | Exacerbation of ulcerative colitis |
|-------------|---------|------------------------------------------------|
| J410. | All | Ulcerative proctocolitis |
| J4100 | All | Ulcerative ileocolitis |
| J410z | All | Ulcerative proctocolitis NOS |
| J4103 | Y30D7 | Ulcerative proctitis |
| Jyu41 | All | [X]Other ulcerative colitis |
| SNOMED Code | Term ID | Description |
| 13470001 | | Chronic ulcerative ileocolitis (disorder) |
| 14311001 | | Severe chronic ulcerative colitis (disorder) |
| 15342002 | | Chronic ulcerative enterocolitis (disorder) |
| 24829000 | | Eosinophilic ulcerative colitis (disorder) |
| 43752006 | | Ulcerative colitis and/or proctitis |
| 52231000 | | Chronic ulcerative proctitis (disorder) |
| 52506002 | | Chronic ulcerative rectosigmoiditis (disorder) |
| 64766004 | | Ulcerative colitis (disorder) |
| 78324009 | | Mild chronic ulcerative colitis (disorder) |
| 78712000 | | Moderate chronic ulcerative colitis (disorder) |
| 128600008 | | Acute ulcerative colitis (disorder) |
| 155764007 | | Ulcerative colitis |
| 196986004 | | Ulcerative proctocolitis |
| 196987008 | | Ulcerative ileocolitis |
| 196988003 | | Ulcerative colitis |
| 196989006 | | Ulcerative proctocolitis |
| 196990002 | | Ulcerative proctocolitis NOS |
| 196991003 | | Ulcerative enterocolitis |
| 196992005 | | Ulcerative ileocolitis |
| 197535008 | | [X]Other ulcerative colitis |
| 201727001 | | Arthropathy in ulcerative colitis (disorder) |

| 201807008 | Juvenile arthritis in ulcerative colitis (disorder) |
|---|---|
| 235714007 | Ulcerative enterocolitis (disorder) |
| 266447004 | Ulcerative colitis |
| 275549008 | History of ulcerative colitis (situation) |
| 295046003 | Ulcerative proctocolitis (disorder) |
| 404908004 | Toxic megacolon due to ulcerative colitis (disorder) |
| 410484008 | Iritis with ulcerative colitis (disorder) |
| 414156000 | Exacerbation of ulcerative colitis (disorder) |
| 441971007 | Chronic left-sided ulcerative colitis (disorder) |
| 442159003 | Chronic ulcerative pancolitis (disorder) |
| 444546002 | Chronic ulcerative colitis (disorder) |
| 444548001 | Ulcerative pancolitis (disorder) |
| 445243001 | Left sided ulcerative colitis (disorder) |
| 697969008 | Ulcerative colitis in remission (disorder) |
| <b>5</b> 22266020 | Secondary autoimmune hemolytic anemia co-occurrent and due to ulcerative |
| 732966008 | colitis (disorder) |
| 1005121000110105 | Abscess of intestine co-occurrent and due to chronic ulcerative pancolitis (disorder) |
| 1085131000119105'<br>1085141000119101' | |
| 1085141000119101 | Complication due to chronic ulcerative pancolitis (disorder) |
| | Fistula of intestine due to chronic ulcerative pancolitis (disorder) |
| 1085161000119102' | Intestinal obstruction due to chronic ulcerative pancolitis (disorder) |
| 1085171000119108' | Rectal hemorrhage due to chronic ulcerative pancolitis (disorder) |
| 1085181000119106' | Abscess of intestine co-occurrent and due to chronic ulcerative proctitis (disorder) |
| 1085191000119109' | Complication due to chronic ulcerative proctitis (disorder) |
| 1085201000119107' | Fistula of intestine due to chronic ulcerative proctitis |
| 1085211000119105' | Intestinal obstruction due to chronic ulcerative proctitis (disorder) |
| 1085221000119103' | Rectal hemorrhage due to chronic ulcerative proctitis |

| | | Abscess of intestine co-occurrent and due to chronic ulcerative rectosigmoiditis |
|---|---|---|
| 1085231000119100' | | (disorder) |
| 1085241000119109' | | Complication due to chronic ulcerative rectosigmoiditis (disorder) |
| 1085251000119106' | | Fistula of large intestine due to chronic ulcerative rectosigmoiditis (disorder) |
| 1085261000119108' | | Intestinal obstruction due to chronic ulcerative rectosigmoiditis (disorder) |
| 1085271000119102' | | Rectal hemorrhage due to chronic ulcerative rectosigmoiditis (disorder) |
| 1092841000119100' | | Abscess of intestine co-occurrent and due to ulcerative colitis (disorder) |
| 1092851000119103' | | Complication due to ulcerative colitis (disorder) |
| 1092861000119101' | | Fistula of intestine due to ulcerative colitis (disorder) |
| 1092871000119107' | | Intestinal obstruction due to ulcerative colitis (disorder) |
| 1092881000119105' | | Rectal hemorrhage due to ulcerative colitis (disorder) |
| Crohn's Disease (CD) | | |
| Read V2 Code | Term ID | Description |
| J40 | All | Regional enteritis- Crohn's disease |
| J400. | All | Regional enteritis of the small bowel |
| J4000 | All | Regional enteritis of the duodenum |
| J4001 | All | Regional enteritis of the jejunum |
| J4002 | All | Crohn's disease of the termnal ileum |
| J4003 | All | Crohn's disease of the ileum unspecified |
| J4004 | All | Crohn's disease of the ileum NOS |
| J4005 | All | Exacerbation of Crohn's disease of small intestine |
| J400z | All | Crohn's disease of the small bowel NOS |
| J4010 | All | Regional enteritis of the colon |
| J4011 | All | Regional enteritis of the rectum |
| J4012 | All | Exacerbation of Crohn's disease of large intestine |
| J401z | All | Crohn's disease of the largel bowel NOS |
| J40z. | All | Crohn's disease NOS |
| Read CTV3 Code | Term ID | Description |

| XE2QL | All | Crohn's disease |
|-------------|---------|----------------------------------------------------|
| Xa0lh | All | Regional enteritis |
| X302r | All | Crohn's jejunitis |
| X302t | All | Crohn's ileitis |
| J4003 | All | Crohn's disease of the ileum unspecified |
| J4004 | All | Crohn's disease of the ileum NOS |
| J4002 | All | Crohn's disease of terminal ileum |
| J400. | All | Regional enteritis of small bowel |
| XaK6C | All | Exacerbation of Crohn's disease of small intestine |
| J400z | All | Crohn's disease of the small bowel NOS |
| J401. | All | Regional enteritis of the large bowel |
| XE0af | All | Crohn's disease of the large bowel NOS |
| XaK6D | All | Exacerbation of Crohn's disease of large intestine |
| J40z. | All | Regional enteritis NOS |
| J4010 | All | Crohn's colitis |
| J4011 | All | Crohn's proctitis |
| X3050 | All | Perianal Crohn's disease |
| J4001 | Y30Fy | Regional enteritis of the jejunum |
| Jyu40 | All | [X]Other Crohn's disease |
| SNOMED Code | Term ID | Description |
| 3815005 | | Crohn's disease of rectum (disorder) |
| 7620006 | | Crohn's disease of large bowel (disorder) |
| 34000006 | | Crohn's disease (disorder) |
| 38106008 | | Crohn's disease of ileum (disorder) |
| 50440006 | | Crohn's disease of colon (disorder) |
| 56287005 | | Crohn's disease of duodenum (disorder) |
| 56689002 | | Crohn's disease of small intestine (disorder) |
| 61424003 | | Crohn's disease of pylorus (disorder) |

| 70622003 | Crohn's disease of pyloric antrum (disorder) |
|-----------|---------------------------------------------------------------|
| 71833008 | Crohn's disease of small AND large intestines (disorder) |
| 91390005 | Crohn's disease of jejunum (disorder) |
| 155761004 | Regional enteritis of small bowel |
| 155762006 | Regional enteritis of the large bowel |
| 155763001 | Regional enteritis NOS |
| 196578009 | Crohn's disease of oral soft tissues (disorder) |
| 196975001 | Regional enteritis - Crohn's disease |
| 196976000 | Regional enteritis of the jejunum |
| 196977009 | Crohn's disease of terminal ileum (disorder) |
| 196978004 | Crohn's disease of the ileum unspecified |
| 196979007 | Crohn's disease of the ileum NOS |
| 196980005 | Crohn's disease of the small bowel NOS |
| 196981009 | Regional enteritis of the large bowel |
| 196982002 | (Crohn's colitis) or (Crohn's disease of the large bowel NOS) |
| 197534007 | [X]Other Crohn's disease |
| 201728006 | Arthropathy in Crohn's disease (disorder) |
| 201805000 | Juvenile arthritis in Crohn's disease (disorder) |
| 234999001 | Crohn's disease of gingivae (disorder) |
| 235607002 | Crohn's disease of esophagus (disorder) |
| 235664007 | Crohn's disease of stomach (disorder) |
| 235796008 | Perianal Crohn's disease (disorder) |
| 266446008 | Crohn's disease of the large bowel NOS |
| 266517004 | Regional enteritis - Crohn |
| 273364009 | Crohn's disease activity index (assessment scale_ |
| 278522007 | Regional enteritis |
| 397172008 | Gastrointestinal Crohn's disease (disorder) |
| 397173003 | Crohn's disease of intestine (disorder) |

| 399946006 | Crohn's disease of skin (disorder) |
|---|---|
| 402375009 | Crohn's disease of vulva (disorder) |
| 402376005 | Crohn's disease of penis (disorder) |
| 402377001 | Crohn's disease of scrotum (disorder) |
| 402378006 | Metastatic Crohn's disease of skin (disorder) |
| 410485009 | Iritis with Crohn's disease (disorder) |
| 413276006 | Crohn's stricture of colon (disorder) |
| 414153008 | Exacerbation of Crohn's disease of large intestine (disorder) |
| 414154002 | Exacerbation of Crohn's disease of small intestine (disorder) |
| 426549001 | Crohn's disease in remission (disorder) |
| 721702009 | Crohn disease of anal canal (disorder) |
| 722850002 | Crohn's disease of gastrointestinal anastomosis (disorder) |
| 726101009 | Extraintestinal Crohn's (disorder) |
| 733157003 | Crohn disease of appendix (disorder) |
| 733533008 | Perianal fistula due to Crohn's disease (disorder) |
| 737195007 | Crohn disease of upper gastrointestinal tract (disorder) |
| 8161000119106' | Arthritis co-occurrent and due to Crohn's disease (disorder) |
| 112561000119108' | History of Crohns disease (situation) |
| 1085751000119100' | Abscess of intestine co-occurrent and due to Crohn's disease of large intestine (disorder) |
| 1085761000119103' | Complication due to Crohn's disease of large intestine (disorder) |
| 1085771000119109' | Fistula of large intestine due to Crohn's disease (disorder) |
| 1085781000119107' | Intestinal obstruction due to Crohn's disease of large intestine (disorder) |
| 1085791000119105' | Rectal hemorrhage due to Crohn's disease of large intestine (disorder) |
| 1085801000119106' | Abscess of intestine co-occurrent and due to Crohn's disease of small and large intestine (disorder) |
| 1085811000119109' | Complication due to Crohn's disease of small and large intestines (disorder) |
| 1085821000119102' | Fistula of intestine due to Crohn's disease of small and large intestine (disorder) |

| 1085831000119104' | Intestinal obstruction due to Crohn's disease of small and large intestine (disorder) |
|---|---|
| 1085841000119108' | Rectal hemorrhage due to Crohn's disease of small and large intestines (disorder) |
| 1085851000119105' | Abscess of intestine co-occurrent and due to Crohn's disease of small intestine (disorder) |
| 1085861000119107' | Complication due to Crohn's disease of small intestine (disorder) |
| 1085871000119101' | Fistula of small intestine due to Crohn's disease (disorder) |
| 1085881000119103' | Intestinal obstruction due to Crohn's disease of small intestine (disorder) |
| 1085891000119100' | Rectal hemorrhage due to Crohn's disease of small intestine (disorder) |
| 1085901000119101' | Abscess of intestine co-occurrent and due to Crohn's disease (disorder) |
| 1085911000119103' | Complication due to Crohn's disease (disorder) |
| 1085931000119108' | Intestinal obstruction due to Crohn's disease (disorder) |
| 1085941000119104' | Rectal hemorrhage due to Crohn's disease (disorder) |
| 10743231000119101' | Stenosis of small intestine co-occurrent and due to Crohn's disease (disorder) |

| Inflammatory Bowel Disease unclassified (IBDU) | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| J4 | All | Inflammatory bowel disease |
| J402. | All | Regional ileocolitis |
| J41y. | All | Other idiopathic proctocolitis |
| J41y1 | All | Toxic megacolon |
| J41yz | All | Other idiopathic proctocolitis NOS |
| J41z. | All | Idiopathic proctocolitis NOS |
| J43 | All | Other non-infective inflammatory gastroenteritis and colitis |
| J435. | All | Pouchitis |

| J437. | All | Colitis |
|---|---|---|
| J438. | All | Left sided colitis |
| J4z2. | All | Non-infective ileitis NOS |
| J4z3. | All | Non-infective colitis NOS |
| J4z4. | All | Non-infective sigmoiditis NOS |
| J4z5. | All | Exacerbation of non-infective colitis |
| J4z6. | All | Indeterminate colitis |
| Read CTV3 Code | Term ID | Description |
| XE0ae | All | Inflammatory bowel disease |
| J402. | All | Regional ileocolitis |
| X303k | All | Indeterminate colitis |
| J41y1 | All | Toxic megacolon |
| XaB5z | All | Enterocolitis |
| XE0aj | All | Other non-infective inflammatory gastroenteritis and colitis |
| Xa3fm | All | Non-infective gastrointestinal inflammation, NOS |
| XaB5x | All | Non-infective enteritis and colitis |
| XaK6F | All | Exacerbation of non-infective colitis |
| X303f | All | Colitis |
| XaRD4 | All | Eosinophilic colitis |
| X303j | All | Non-Crohn's granulomatous colitis |
| Xa7nY | All | Non-infective colitis |
| J4z3. | All | Non-infective colitis NOS |
| X304G | All | Sigmoiditis |
| J4z4. | All | Non-infective sigmoiditis NOS |
| X3047 | All | Proctitis |
| J574C | All | Proctitis NOS |
| X303e | All | Proctocolitis |
| J41y. | All | Other idiopathic proctocolitis |

| J41yz | All | Other idiopathic proctocolitis NOS |
|---|---|---|
| J41z. | All | Idiopathic proctocolitis NOS |
| X304F | All | Caecitis |
| SNOMED Code | Term ID | Description |
| 24526004 | | Inflammatory bowel disease (disorder) |
| 721686000 | | Inflammatory polyps co-occurrent and due to inflammatory bowel disease (disorder) |
| 6382002 | | Chronic inflammatory small bowel disease (disorder) |
| 771333006 | | Immune dysregulation, inflammatory bowel disease, arthritis, recurrent infection syndrome (disorder) |
| 128999004 | | Inflammatory disorder of digestive tract (disorder) |
| 64226004 | | Colitis |
| 54597004 | | Chronic colitis (disorder) |
| 369445005 | | Chronic proctocolitis (disorder) |
| 369447002 | | Chronic proctocolitis, confluent (disorder) |
| 369446006 | | Chronic proctocolitis, patchy (disorder) |
| 52506002 | | Chronic ulcerative rectosigmoiditis (disorder) |
| 373639002 | | Distal colitis (disorder) |
| 51290000 | | Diversion colitis (disorder) |
| 29120000 | | Eosinophilic colitis (disorder) |
| 783185002 | | Focal active colitis (disorder) |
| 359660000 | | Idiopathic colitis (disorder |
| 235746007 | | Indeterminate colitis (disorder) |
| 43752006 | | Inflammation of small intestine and colon (disorder) |
| 13470001 | | Chronic ulcerative ileocolitis (disorder) |
| 71207007 | | Noninfectious enteritis (disorder) |
| 735731005 | | Chronic non-infectious enteritis of uncertain etiology (disorder) |
| 307418008 | | Non-infective enteritis and colitis (disorder) |
| 14066009 | | Noninfectious colitis (disorder) |

| 414155001 | Exacerbation of non-infective colitis (disorder) |
|-----------|----------------------------------------------------------------|
| 53372009 | Noninfectious sigmoiditis (disorder) |
| 788718000 | Iritis co-occurrent with inflammatory bowel disease (disorder) |
| 64613007 | Inflammation of small intestine (disorder) |
| 52457000 | Ileitis (disorder) |
| 51151007 | Noninfectious ileitis (disorder) |
| 196983007 | Regional ileocolitis (disorder) |
| 302168000 | Inflammation of large intestine (disorder) |
| 3951002 | Proctitis (disorder) |
| 313327004 | Inflammatory cloacogenic polyp (disorder) |
| 28536002 | Toxic megacolon (disorder) |

**sTable 1.2** WHO International Statistical Classification of Diseases (ICD-10) to be used to codes to be used to identify cases of IBD and IBD subtypes

| Clinical entity | ICD 10 code | Definition |
|--------------------|-------------|---------------------------------------|
| Crohn's disease | K50 | Any diagnostic or indicative code for |
| | | Crohn's disease, excluding ulcerative |
| | | colitis |
| Ulcerative colitis | K51 | Any diagnostic or indicative code for |
| | | ulcerative colitis |

# Appendix 2

**sTable 2.1** Read and SNOMED codes to be used to identify mental health conditions

| Depressive episode | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| E112. | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| E1123 | All | Single major depressive episode, severe, without mention of psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E118. | All | Seasonal affective disorder |
| E11y2 | All | Atypical depressive disorder |

| E11z2 | All | Marked depression |
|-------|-----|------------------------------------------------------------|
| | | Masked depression |
| E130. | All | Reactive depressive psychosis |
| E135. | All | Agitated depression |
| E2003 | All | Anxiety with depression |
| E291. | All | Prolonged depressive reaction |
| E2B | All | Depressive disorder NEC |
| E2B1. | All | Chronic depression |
| E2B0. | All | Postviral depression |
| Eu204 | All | [X]Post-schizophrenic depression |
| Eu251 | All | [X]Schizoaffective disorder, depressive type |
| Eu32. | All | [X]Depressive episode |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu322 | All | [X]Severe depressive episode without psychotic symptoms |
| Eu323 | All | [X]Severe depressive episode with psychotic symptoms |
| Eu324 | All | [X]Mild depression |
| Eu325 | All | [X]Major depression, mild |
| Eu326 | All | [X]Major depression, moderately severe |
| Eu327 | All | [X]Major depression, severe without psychotic symptoms |
| Eu328 | All | [X]Major depression, severe with psychotic symptoms |
| Eu32y | All | [X]Other depressive episodes |
| Eu32z | All | [X]Depressive episode, unspecified |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |

| | | [X]Recurrent depressive disorder, current episode severe without psychotic |
|---|---|---|
| Eu332 | All | symptoms |
| | | [X]Recurrent depressive disorder, current episode severe with psychotic |
| Eu333 | All | symptoms |
| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Eu412 | All | [X]Mixed anxiety and depressive disorder |
| Read CTV3 Code | Term ID | Description |
| X00Sb | All | Mixed anxiety and depressive disorder |
| X00SO | All | Depressive disorder |
| X761L | All | Seasonal affective disorder |
| Xa0wV | All | Recurrent brief depressive disorder |
| X00SQ | All | Agitated depression |
| XE1YC | All | Reactive depression |
| X00SR | All | Endogenous depression |
| X00SS | All | Endogenous depression first episode |
| XE1Y0 | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| E1123 | All | Single major depressive episode, severe, without mention of psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| XaX53 | All | Single major depressive episode, severe, with psychosis, psychosis in remission |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |

| XM1GC | All | Endogenous depression - recurrent |
|---|---|---|
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |
| X00SU | All | Masked depression |
| E11y2 | All | Atypical depressive disorder |
| X00S8 | All | Post-schizophrenic depression |
| XSEGJ | All | Major depressive disorder |
| XSKr7 | All | Cotard syndrome |
| XSGol | All | Moderate major depression |
| XSGok | All | Mild major depression |
| XSGom | All | Severe major depression without psychotic features |
| XSGon | All | Severe major depression with psychotic features |
| E1137 | All | Recurrent depression |
| E130. | All | Reactive depressive psychosis |
| E2B | All | Depressive disorder NEC |
| E2B0. | All | Postviral depression |
| E2B1. | All | Chronic depression |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |

| XE1Y1 | All | Recurrent major depressive episodes |
|---|---|---|
| XE1ZY | All | [X]Severe depressive episode without psychotic symptoms |
| XE1ZZ | All | [X]Severe depressive episode with psychotic symptoms |
| XE1Za | All | [X]Other depressive episodes |
| XE1Zb | All | [X]Depressive episode, unspecified |
| | | [X]Recurrent depressive disorder, current episode severe without psychotic |
| XE1Zd | All | symptoms |
| | | [X]Recurrent depressive disorder, current episode severe with psychotic |
| XE1Ze | All | symptoms |
| XE1Zf | All | [X]Recurrent depressive disorder, unspecified |
| XaB9J | All | Depression NOS |
| XaCHr | All | [X] Single episode agitated depression without psychotic symptoms |
| XaCHs | All | [X] Single episode major depression without psychotic symptoms |
| XaCIs | All | Mild depression |
| XaCIt | All | Moderate depression |
| XaCIu | All | Severe depression |
| SNOMED Code | Term ID | Description |
| 832007' | | Moderate major depression (disorder) |
| 2618002' | | Chronic recurrent major depressive disorder (disorder) |
| 14070001' | | Multi-infarct dementia with depression (disorder) |
| 14183003' | | Chronic major depressive disorder, single episode (disorder) |
| | | Severe recurrent major depression with psychotic features, mood-incongruent |
| 15193003' | | (disorder) |
| 15639000' | | Moderate major depression, single episode (disorder) |
| 18818009' | | Moderate recurrent major depression (disorder) |
| 19527009' | | Single episode of major depression in full remission (disorder) |

| | Seve | ere major depression, single episode, with psychotic features, mood- |
|---|---|---|
| 20250007' | inco | ngruent (disorder) |
| 25922000' | Majo | or depressive disorder, single episode with postpartum onset (disorder) |
| 28475009' | Seve | ere recurrent major depression with psychotic features (disorder) |
| 30605009' | Majo | or depression in partial remission (disorder) |
| 33078009' | | ere recurrent major depression with psychotic features, mood-congruent order) |
| 33135002' | Reci | urrent major depression in partial remission (disorder) |
| 33736005' | Seve | ere major depression with psychotic features, mood-congruent (disorder) |
| 35489007' | Dep | ressive disorder (disorder) |
| 36474008' | Seve | ere recurrent major depression without psychotic features (disorder) |
| 36923009' | Majo | or depression, single episode (disorder) |
| 38694004' | Reci | urrent major depressive disorder with atypical features (disorder) |
| 39809009' | Reci | urrent major depressive disorder with catatonic features (disorder) |
| 40379007' | Mild | l recurrent major depression (disorder) |
| 40568001' | Recu | urrent brief depressive disorder (disorder) |
| 42925002' | Majo | or depressive disorder, single episode with atypical features (disorder) |
| 48589009' | Min | or depressive disorder (disorder) |
| 58703003' | Post | partum depression (disorder) |
| 60099002' | Seve | ere major depression with psychotic features, mood-incongruent (disorder) |
| 66344007' | Reci | urrent major depression (disorder) |
| 69392006' | Majo | or depressive disorder, single episode with catatonic features (disorder) |
| 70747007' | Majo | or depression single episode, in partial remission (disorder) |
| 71336009' | Recu | urrent major depressive disorder with postpartum onset (disorder) |
| 73867007' | Seve | ere major depression with psychotic features (disorder) |
| 75084000' | Seve | ere major depression without psychotic features (disorder) |
| 76441001' | Seve | ere major depression, single episode, without psychotic features (disorder) |

| | Severe major depression, single episode, with psychotic features, mood- |
|---|---|
| 77911002' | congruent (disorder) |
| 79298009' | Mild major depression, single episode (disorder) |
| 79842004' | Stuporous depression (disorder) |
| 82218004' | Postoperative depression (disorder) |
| 83458005' | Agitated depression (disorder) |
| 87414006' | Reactive depression (situational) (disorder) |
| 87512008' | Mild major depression (disorder) |
| 161469008' | History of depression (situation) |
| 191466007' | Arteriosclerotic dementia with depression (disorder) |
| 191495003' | Drug-induced depressive state (disorder) |
| 191604000' | Single major depressive episode, severe, with psychosis (disorder) |
| 191610000' | Recurrent major depressive episodes, mild (disorder) |
| 191611001' | Recurrent major depressive episodes, moderate (disorder) |
| 191613003' | Recurrent major depressive episodes, severe, with psychosis (disorder) |
| 191616006' | Recurrent depression (disorder) |
| 191659001' | Atypical depressive disorder (disorder) |
| 191676002' | Reactive depressive psychosis (disorder) |
| 192046006' | Brief depressive adjustment reaction (disorder) |
| 192049004' | Prolonged depressive adjustment reaction (disorder) |
| 192079006' | Postviral depression (disorder) |
| 192080009' | Chronic depression (disorder) |
| 231485007' | Post-schizophrenic depression (disorder) |
| 231499006' | Endogenous depression first episode (disorder) |
| 231500002' | Masked depression (disorder) |
| 231504006' | Mixed anxiety and depressive disorder (disorder) |

| 237349002' | Mild postnatal depression (disorder) |
|---|---|
| 237350002' | Severe postnatal depression (disorder) |
| 237739002' | Pseudo-Cushing's syndrome of depression (disorder) |
| 247803002' | Seasonal affective disorder (disorder) |
| 268621008' | Recurrent major depressive episodes (disorder) |
| 272022009' | Complaining of feeling depressed (finding) |
| 274948002' | Endogenous depression - recurrent (disorder) |
| 300706003' | Endogenous depression (disorder) |
| 310495003' | Mild depression (disorder) |
| 310496002' | Moderate depression (disorder) |
| 310497006' | Severe depression (disorder) |
| 319768000' | Recurrent major depressive disorder with melancholic features (disorder) |
| 320751009' | Major depression, melancholic type (disorder) |
| 321717001' | Involutional depression (disorder) |
| 366979004' | Depressed mood (finding) |
| 370143000' | Major depressive disorder (disorder) |
| 394924000' | Symptoms of depression (finding) |
| 395072006' | Counseling for postnatal depression (procedure) |
| 430852001' | Severe major depression, single episode, with psychotic features (disorder) |
| 450714000' | Severe major depression (disorder) |
| 704678007' | Depressed mood with postpartum onset (finding) |
| 712823008' | Acute depression (disorder) |
| 718636001' | Minimal depression (disorder) |
| 719592004' | Moderately severe major depression (disorder) |
| 719593009' | Moderately severe depression (disorder) |
| 720451004' | Minimal recurrent major depression (disorder) |

| 720452006' | Moderately severe recurrent major depression (disorder) |
|---|---|
| 720453001' | Moderately severe major depression single episode (disorder) |
| 720454007' | Minimal major depression single episode (disorder) |
| 720455008' | Minimal major depression (disorder) |
| 723928009' | Mood disorder with depressive symptoms caused by alcohol (disorder) |
| | Mood disorder with mixed manic and depressive symptoms caused by alcohol |
| 723930006' | (disorder) |
| 724676000' | Mood disorder with depressive symptoms caused by sedative (disorder) |
| 724677009' | Mood disorder with depressive symptoms caused by hypnotic (disorder) |
| 724678004' | Mood disorder with depressive symptoms caused by anxiolytic (disorder) |
| 724690002' | Mood disorder with depressive symptoms caused by cocaine (disorder) |
| 724757005' | Depressive symptoms due to primary psychotic disorder (disorder) |
| 726772006' | Major depression with psychotic features (disorder) |
| 762321000' | Mood disorder with depressive symptoms caused by opioid (disorder) |
| 762329003' | Mood disorder with depressive symptoms caused by stimulant (disorder) |
| 762336002' | Mood disorder with depressive symptoms caused by hallucinogen (disorder) |
| 762339009' | Mood disorder with depressive symptoms caused by volatile inhalant (disorder) |
| | Mood disorder with depressive symptoms caused by synthetic cathinone |
| 762512002' | (disorder) |
| 768835002' | Depression care management (procedure) |
| 788120007' | Antenatal depression (disorder) |
| | Mood disorder with mixed depressive and manic symptoms caused by |
| 838529004' | amfetamine and amfetamine derivative (disorder) |
| 871840004' | Episode of depression (finding) |
| 251000119105' | Severe major depression, single episode (disorder) |
| 281000119103' | Severe recurrent major depression (disorder) |
| 10211000132109' | Perinatal depression (disorder) |
| 94631000119100' | Depressive disorder in mother complicating pregnancy (disorder) |
|---|---|
| 133121000119109' | Severe seasonal affective disorder (disorder) |
| 199111000000100' | Referral for guided self-help for depression (procedure) |
| 286711000000107' | Counseling for depression (procedure) |
| 288751000119101' | Reactive depressive psychosis, single episode (disorder) |
| 361761000000106' | On full dose long term treatment for depression (finding) |
| 755321000000106' | Single major depressive episode, severe, with psychosis, psychosis in remission (disorder) |
| 755331000000108' | Recurrent major depressive episodes, severe, with psychosis, psychosis in remission (disorder) |
| 764611000000100' | Recurrent major depressive episodes, severe (disorder) |
| 764691000000109' | Recurrent major depressive episodes, in partial remission (disorder) |
| 764701000000109' | Recurrent major depressive episodes, in remission (disorder) |
| 764711000000106' | Single major depressive episode, in remission (disorder) |
| 923921000000104' | Referral for depression self-help video (procedure) |
| 1086471000000100' | Recurrent reactive depressive episodes, severe, with psychosis (disorder) |
| 1086661000000100' | Reactive depression, prolonged single episode (disorder) |
| 1086671000000100' | Reactive depression, single episode (disorder) |
| 1086681000000100' | Reactive depression, recurrent (disorder) |
| 1086691000000100' | Reactive depression, first episode (disorder) |
| 1089511000000100' | Recurrent depression with current severe episode and psychotic features (disorder) |
| | Recurrent depression with current severe episode without psychotic features |
| 1089631000000100' | (disorder) |
| 1089641000000100' | Recurrent depression with current moderate episode (disorder) |
| 10811121000119100' | Major depressive disorder in mother complicating childbirth (disorder) |
| 10811161000119100' | Major depressive disorder in mother complicating pregnancy (disorder) |

| 10835871000119100' | | Depressive disorder in mother complicating childbirth (disorder) |
|---|---|---|
| 16238181000119100' | | Depressive disorder caused by amphetamine (disorder) |
| 16238221000119100' | | Depressive disorder caused by methamphetamine (disorder) |
| 16264621000119100' | | Recurrent mild major depressive disorder co-occurrent with anxiety (disorder) |
| 16264821000119100' | | Recurrent severe major depressive disorder co-occurrent with anxiety (disorder) |
| | | Recurrent moderate major depressive disorder co-occurrent with anxiety |
| 16264901000119100' | | (disorder) |
| | | Recurrent major depressive disorder in partial remission co-occurrent with |
| 16265301000119100' | | anxiety (disorder) |
| | | Mild major depressive disorder co-occurrent with anxiety single episode |
| 16265951000119100' | | (disorder) |
| | | Moderate major depressive disorder co-occurrent with anxiety single episode |
| 16266831000119100' | | (disorder) |
| | | Severe major depressive disorder co-occurrent with anxiety single episode |
| 16266991000119100' | | (disorder) |
| Anxiety episode | | |
| Read V2 Code | Term ID | Description |
| E200. | All | Anxiety states |
| E2000 | All | Anxiety state unspecified |
| E2001 | All | Panic disorder |
| E2002 | All | Generalised anxiety disorder |
| E2003 | All | Anxiety with depression |
| E2004 | All | Chronic anxiety |
| E2005 | All | Recurrent anxiety |
| E200z | All | Anxiety state NOS |
| Eu41. | All | [X]Other anxiety disorders |
| Eu410 | All | [X]Panic disorder [episodic paroxysmal anxiety] |

| Eu411 | All | [X]Generalized anxiety disorder |
|---|---|---|
| Eu412 | All | [X]Mixed anxiety and depressive disorder |
| Eu413 | All | [X]Other mixed anxiety disorders |
| Eu41y | All | [X]Other specified anxiety disorders |
| Eu41z | All | [X]Anxiety disorder, unspecified |
| Read CTV3 Code | Term ID | Description |
| E200. | All | Anxiety disorder |
| XE1Y7 | All | Panic disorder |
| Eu410 | All | [X]Panic disorder [episodic paroxysmal anxiety] |
| E2002 | All | Generalised anxiety disorder |
| X00Sb | All | Mixed anxiety and depressive disorder |
| X00RP | All | Organic anxiety disorder |
| E2004 | All | Chronic anxiety |
| E2005 | All | Recurrent anxiety |
| E200z | All | Anxiety state NOS |
| X00Sc | All | Anxiety hysteria |
| Eu41. | All | [X]Other anxiety disorders |
| Eu413 | All | [X]Other mixed anxiety disorders |
| Eu41z | All | [X]Anxiety disorder, unspecified |
| XE1Zj | All | [X]Other specified anxiety disorders |
| SNOMED Code | Term ID | Description |
| 1037451000000100' | | Referral for psychological management of anxiety (procedure) |
| 1053831000000100' | | Signposting to Anxiety UK (procedure) |
| 10586006' | | Occupation-related stress disorder (disorder) |
| 10743001000119100' | | Anxiety disorder in mother complicating childbirth (disorder) |
| 109006' | | Anxiety disorder of childhood OR adolescence (disorder) |

| 111487009' | Dream anxiety disorder (disorder) |
|---|---|
| 11458009' | Anticipatory anxiety, mild (finding) |
| 11806006' | Separation anxiety disorder of childhood (disorder) |
| 12398201000119100' | Anxiety disorder caused by methamphetamine (disorder) |
| 126943008' | Separation anxiety (disorder) |
| 13438001' | Overanxious disorder of childhood (disorder) |
| 15277004' | Hallucinogen-induced anxiety disorder (disorder) |
| 161470009' | History of anxiety state (situation) |
| 16264621000119100' | Recurrent mild major depressive disorder co-occurrent with anxiety (disorder) |
| 16264821000119100' | Recurrent severe major depressive disorder co-occurrent with anxiety (disorder) |
| 16264901000119100' | Recurrent moderate major depressive disorder co-occurrent with anxiety |
| | (disorder) |
| 16265301000119100' | Recurrent major depressive disorder in partial remission co-occurrent with |
| | anxiety (disorder) |
| 16265701000119100' | Illness anxiety disorder (disorder) |
| 16265951000119100' | Mild major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266831000119100' | Moderate major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266991000119100' | Severe major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 162723006' | On examination - anxious (finding) |
| 1686006' | Sedative, hypnotic AND/OR anxiolytic-induced anxiety disorder (disorder) |
| 17496003' | Organic anxiety disorder (disorder) |
| 191708009' | Chronic anxiety (finding) |
| 191709001' | Recurrent anxiety (finding) |
| 192108001' | Disturbance of anxiety and fearfulness in childhood and adolescence (disorder) |

| 192611004' | Childhood phobic anxiety disorder (disorder) |
|------------------|--------------------------------------------------|
| 197480006' | Anxiety disorder (disorder) |
| 198288003' | Anxiety state (finding) |
| 207363009' | Anxiety neurosis (finding) |
| 21897009' | Generalized anxiety disorder (disorder) |
| 225216003' | Acknowledging anxiety (procedure) |
| 225624000' | Panic attack (finding) |
| 22621000119103' | Anxiety disorder caused by drug (disorder) |
| 228560001' | Anxiety management training (procedure) |
| 231502005' | Situational panic attack (finding) |
| 231503000' | Non-situational panic attack (finding) |
| 231504006' | Mixed anxiety and depressive disorder (disorder) |
| 231506008' | Anxiety hysteria (finding) |
| 247805009' | Anxiety and fear (finding) |
| 286644009' | Level of anxiety (finding) |
| 286710008' | Anxious character (finding) |
| 286711007' | Over-anxious character (finding) |
| 286712000' | Fearful character (finding) |
| 300895004' | Anxiety attack (finding) |
| 313087008' | Counseling for anxiety (procedure) |
| 34938008' | Alcohol-induced anxiety disorder (disorder) |
| 351861000000106' | Stranger anxiety (disorder) |
| 35429005' | Anticipatory anxiety (finding) |
| 35607004' | Panic disorder with agoraphobia (disorder) |
| 36646009' | Anticipatory anxiety, moderate (finding) |
| 371631005' | Panic disorder (disorder) |

| 37868008' | Anxiety disorder of adolescence (disorder) |
|---|---|
| 37872007' | Avoidant disorder of childhood OR adolescence (disorder) |
| 386808001' | Phobia (finding) |
| 386810004' | Phobic anxiety disorder (disorder) |
| 395017009' | Complaining of panic attack (finding) |
| 405051006' | Level of anxiety (observable entity) |
| 417676004' | On examination - panic attack (finding) |
| 43150009' | Panic disorder without agoraphobia with severe panic attacks (disorder) |
| 47372000' | Adjustment disorder with anxious mood (disorder) |
| 48694002' | Anxiety (finding) |
| 50026000' | Psychoactive substance-induced organic anxiety disorder (disorder) |
| 51493001' | Cocaine-induced anxiety disorder (disorder) |
| 51916003' | Biofeedback training by electroencephalogram application in anxiety |
| | (regime/therapy) |
| 52910006' | Anxiety disorder due to a general medical condition (disorder) |
| 53467004' | Anxiety disorder of childhood (disorder) |
| 53956006' | Panic disorder without agoraphobia with panic attacks in partial remission |
| | (disorder) |
| 5509004' | Panic disorder with agoraphobia AND severe panic attacks (disorder) |
| 55967005' | Phencyclidine-induced anxiety disorder (disorder) |
| 56576003' | Panic disorder without agoraphobia (disorder) |
| 5874002' | Anticipatory anxiety, severe (finding) |
| 61387006' | Moderate anxiety (finding) |
| 63909006' | Panic disorder with agoraphobia AND panic attacks in partial remission |
| | (disorder) |
| 64165008' | Avoidant disorder of childhood (disorder) |
| 65064003' | Panic disorder without agoraphobia with moderate panic attacks (disorder) |

| 69479009' | | Anxiety hyperventilation (disorder) |
|---|---|---|
| 70997004' | | Mild anxiety (finding) |
| 710060004' | | Management of anxiety (procedure) |
| 710841007' | | Assessment of anxiety (procedure) |
| 724708007' | | Anxiety disorder caused by methylenedioxymethamphetamine (disorder) |
| 724722007' | | Anxiety disorder caused by dissociative drug (disorder) |
| 724723002' | | Anxiety disorder caused by ketamine (disorder) |
| 72861004' | | Panic disorder without agoraphobia with mild panic attacks (disorder) |
| 737341006' | | Anxiety disorder caused by synthetic cannabinoid (disorder) |
| 762331007' | | Anxiety disorder caused by stimulant (disorder) |
| 788866004' | | Anxiety due to dementia (finding) |
| 80583007' | | Severe anxiety (panic) (finding) |
| 81350009' | | Free-floating anxiety (finding) |
| 8185002' | | Panic disorder with agoraphobia AND moderate panic attacks (disorder) |
| 82339009' | | Amphetamine-induced anxiety disorder (disorder) |
| 85061001' | | Separation anxiety disorder of childhood, early onset (disorder) |
| 858991000000101' | | Provision of written information about generalised anxiety disorder (procedure) |
| 859891000000103' | | Able to manage anxiety (finding) |
| 861611000000100' | | Education about anxiety (procedure) |
| 89948007' | | Panic disorder with agoraphobia AND mild panic attacks (disorder) |
| 90790003' | | Avoidant disorder of adolescence (disorder) |
| 94641000119109' | | Anxiety in pregnancy (disorder) |
| Eating disorders | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |

| Body image disorders | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Attention-deficit disorder (ADHI | 0) | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Behavioural disorders | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Adjustment disorder | | |
| Read V2 Code | Term ID | Description |
| E29 | All | Adjustment reaction |
| E290. | All | Brief depressive reaction |
| E2900 | All | Grief reaction |
| E290z | All | Brief depressive reaction NOS |
| E291. | All | Prolonged depressive reaction |
| E292. | All | Adjustment reaction with predominant disturbance of other emotions |
| E2924 | All | Adjustment reaction with anxious mood |
| E292y | All | Adjustment reaction with mixed disturbance of emotion |
| E292z | All | Adjustment reaction with disturbance of other emotion NOS |
| E293. | All | Adjustment reaction with predominant disturbance of conduct |
| E2930 | All | Adjustment reaction with aggression |
| | | Adjustment reaction with antisocial behaviour |

| E2932 | All | Adjustment reaction with destructiveness |
|---|---|---|
| E293z | All | Adjustment reaction with predominant disturbance of conduct NOS |
| E294. | All | Adjustment reaction with mixed disturbance of emotion and conduct |
| E29y. | All | Other adjustment reactions |
| E29y2 | All | Adjustment reaction with physical symptoms |
| E29y3 | All | Elective mutism due to an adjustment reaction |
| E29y5 | All | Other adjustment reaction with withdrawal |
| E29yz | All | Other adjustment reactions NOS |
| E29z. | All | Adjustment reaction NOS |
| Read CTV3 Code | Term ID | Description |
| E29 | All | Adjustment disorder |
| E290. | All | Brief depressive adjustment reaction |
| E290z | All | Brief depressive reaction NOS |
| E291. | All | Prolonged depressive adjustment reaction |
| E2924 | All | Adjustment reaction with anxious mood |
| E292y | All | Adjustment reaction with mixed disturbance of emotion |
| E293. | All | Adjustment reaction with predominant disturbance of conduct |
| E2930 | All | Adjustment reaction with aggression |
| E2931 | All | Adjustment reaction with antisocial behaviour |
| E2932 | All | Adjustment reaction with destructiveness |
| E293z | All | Adjustment reaction with predominant disturbance of conduct NOS |
| E294. | All | Adjustment reaction with mixed disturbance of emotion and conduct |
| E292. | All | Adjustment reaction with predominant disturbance of other emotions |
| E292z | All | Adjustment reaction with disturbance of other emotion NOS |
| E29y. | All | Other adjustment reactions |
| E29yz | All | Other adjustment reactions NOS |

| E29y2 | All | Adjustment reaction with physical symptoms |
|---|---|---|
| E29y3 | All | Elective mutism due to an adjustment reaction |
| E29y5 | All | Other adjustment reaction with withdrawal |
| E29z. | All | Adjustment reaction NOS |
| SNOMED Code | Term ID | Description |
| 17226007 | | Adjustment disorder (disorder) |
| 15977008 | | Adjustment disorder with academic inhibition (disorder) |
| 47372000 | | Adjustment disorder with anxious mood (disorder) |
| 57194009 | | Adjustment disorder with depressed mood (disorder) |
| 192046006 | | Brief depressive adjustment reaction (disorder) |
| 192049004 | | Prolonged depressive adjustment reaction (disorder) |
| 84984002 | | Adjustment disorder with disturbance of conduct (disorder) |
| 66381006 | | Adjustment disorder with mixed disturbance of emotions AND conduct (disorder) |
| 192056005 | | Adjustment reaction with aggression (disorder) |
| 192057001 | | Adjustment reaction with antisocial behavior (disorder) |
| 192058006 | | Adjustment reaction with destructiveness (disorder) |
| 55668003 | | Adjustment disorder with mixed emotional features (disorder) |
| 18478005 | | Adjustment disorder with physical complaints (disorder) |
| 9674006 | | Adjustment disorder with withdrawal (disorder) |
| 32880007 | | Adjustment disorder with work inhibition (disorder) |
| 386821008 | | Adjustment reaction in infancy (disorder) |
| 386822001 | | Adjustment reaction of adolescence (disorder) |
| 386823006 | | Adjustment reaction of adult life (disorder) |
| 386824000 | | Adjustment reaction of childhood (disorder) |

| 386825004 | | Adjustment reaction of late life (disorder) |
|---|---|---|
| 425914008 | | Adjustment reaction to medical therapy (disorder) |
| 192063005 | | Adjustment reaction with physical symptoms (disorder) |
| 192064004 | | Elective mutism due to an adjustment reaction (disorder) |
| | | Adjustment disorder with mixed disturbance of emotions and conduct in |
| 698697003 | | remission (disorder) |
| Acute stress disorder | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Schizophrenia | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Post-traumatic stress disorder | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Bipolar disorder | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |

**sTable 2.2** Algorithms used to identify anxiety episodes, depression episodes, and recurrent major depression. Expressions in capitals equate to Boolean expressions. \*More than 1 year ago. SSRIs = selective serotonin reuptake inhibitors, TCA = tricyclic antidepressants, MAOI = monoamine oxidase inhibitors, CBT = cognitive behavioural therapy.

| Clinical entity | Definition |
|---------------------|-------------------------------------------|
| Anxiety | Any coded anxiety episode AND concurrent |
| | treatment for anxiety |
| Depressive episode | Any coded depressive episode AND |
| | concurrent treatment for depression |
| Recurrent | (Any historical code* for a depressive |
| depressive disorder | episode AND current treatment for |
| | depression) OR Any code for recurrent |
| | depressive disorder |
| Anxiety treatments | SSRIs, anxiolytics, counselling, CBT, and |
| | psychotherapy |
| Depression | SSRIs, TCAs, MAOIs, counselling, CBT, and |
| treatments | psychotherapy |

**sTable 2.3** WHO International Statistical Classification of Diseases (ICD-10) for mental health conditions

| Clinical entity | ICD 10 code | Definition |
|------------------|-------------|-------------------------------------------|
| Depressive | F32 | Any coded depressive episode AND |
| episode | | concurrent treatment for depression |
| Recurrent | F33 | (Any historical code* for a depressive |
| depressive | | episode AND current treatment for |
| disorder | | depression) OR Any code for recurrent |
| | | depressive disorder |
| Depression | NA | SSRIs, TCAs, MAOIs, counselling, CBT, |
| treatments | | and psychotherapy |
| Anxiety | F41 | Any coded anxiety episode AND |
| | | concurrent treatment for anxiety |
| Anxiety | NA | SSRIs, anxiolytics, counselling, CBT, and |
| treatments | | psychotherapy |
| Self-harm | X60-X84 | Any diagnostic or indicative code for |
| | | any form of self-harm, |
| | | including suicide attempt |
| Eating disorders | F50 | Any diagnostic or indicative code for |
| | | eating disorders |

| Body image | F45.2 | Any diagnostic or indicative code for |
|-------------------|-------|---------------------------------------|
| disorders | | body image / dysmorphic disorder |
| | | (excluding hypochondriacal disorders |
| | | not associated with body image) |
| Attention-deficit | F90.0 | Any diagnostic or indicative code for |
| disorders | | disturbance of activity and attention |
| Behavioural | F91 | Any diagnostic or indicative code for |
| disorders | F92 | conduct disorders |
| Adjustment | F43.2 | Any diagnostic or indicative code for |
| disorders | | adjustment disorders |
| Acute stress | F43.0 | Any diagnostic or indicative code for |
| disorders | | acute stress disorders |
| Post-traumatic | F43.1 | Any diagnostic or indicative code for |
| stress disorder | | Post-traumatic stress disorder |

## Appendix 3

**sTable 3.1** Read and SNOMED codes to be used to identify quality of life

| Depressive episode | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| E112. | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| E1123 | All | Single major depressive episode, severe, without mention of psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E118. | All | Seasonal affective disorder |
| E11y2 | All | Atypical depressive disorder |
| E11z2 | All | Masked depression |
| E130. | All | Reactive depressive psychosis |

| E135. | All | Agitated depression |
|---|---|---|
| E2003 | All | Anxiety with depression |
| E291. | All | Prolonged depressive reaction |
| E2B | All | Depressive disorder NEC |
| E2B1. | All | Chronic depression |
| E2B0. | All | Postviral depression |
| Eu204 | All | [X]Post-schizophrenic depression |
| Eu251 | All | [X]Schizoaffective disorder, depressive type |
| Eu32. | All | [X]Depressive episode |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu322 | All | [X]Severe depressive episode without psychotic symptoms |
| Eu323 | All | [X]Severe depressive episode with psychotic symptoms |
| Eu324 | All | [X]Mild depression |
| Eu325 | All | [X]Major depression, mild |
| Eu326 | All | [X]Major depression, moderately severe |
| Eu327 | All | [X]Major depression, severe without psychotic symptoms |
| Eu328 | All | [X]Major depression, severe with psychotic symptoms |
| Eu32y | All | [X]Other depressive episodes |
| Eu32z | All | [X]Depressive episode, unspecified |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| | | [X]Recurrent depressive disorder, current episode severe without psychotic |
| Eu332 | All | symptoms |
| | | [X]Recurrent depressive disorder, current episode severe with psychotic |
| Eu333 | All | symptoms |

| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
|---|---|---|
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Eu412 | All | [X]Mixed anxiety and depressive disorder |
| Read CTV3 Code | Term ID | Description |
| X00Sb | All | Mixed anxiety and depressive disorder |
| X00SO | All | Depressive disorder |
| X761L | All | Seasonal affective disorder |
| Xa0wV | All | Recurrent brief depressive disorder |
| X00SQ | All | Agitated depression |
| XE1YC | All | Reactive depression |
| X00SR | All | Endogenous depression |
| X00SS | All | Endogenous depression first episode |
| XE1Y0 | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| E1123 | All | Single major depressive episode, severe, without mention of psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| XaX53 | All | Single major depressive episode, severe, with psychosis, psychosis in remission |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| XM1GC | All | Endogenous depression - recurrent |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |

| E1132 | All | Recurrent major depressive episodes, moderate |
|---|---|---|
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |
| X00SU | All | Masked depression |
| E11y2 | All | Atypical depressive disorder |
| X00S8 | All | Post-schizophrenic depression |
| XSEGJ | All | Major depressive disorder |
| XSKr7 | All | Cotard syndrome |
| XSGol | All | Moderate major depression |
| XSGok | All | Mild major depression |
| XSGom | All | Severe major depression without psychotic features |
| XSGon | All | Severe major depression with psychotic features |
| E1137 | All | Recurrent depression |
| E130. | All | Reactive depressive psychosis |
| E2B | All | Depressive disorder NEC |
| E2B0. | All | Postviral depression |
| E2B1. | All | Chronic depression |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| XE1Y1 | All | Recurrent major depressive episodes |
| XE1ZY | All | [X]Severe depressive episode without psychotic symptoms |
| XE1ZZ | All | [X]Severe depressive episode with psychotic symptoms |

| XE1Za | All | [X]Other depressive episodes |
|---|---|---|
| XE1Zb | All | [X]Depressive episode, unspecified |
| | | [X]Recurrent depressive disorder, current episode severe without psychotic |
| XE1Zd | All | symptoms |
| | | [X]Recurrent depressive disorder, current episode severe with psychotic |
| XE1Ze | All | symptoms |
| XE1Zf | All | [X]Recurrent depressive disorder, unspecified |
| XaB9J | All | Depression NOS |
| XaCHr | All | [X] Single episode agitated depression without psychotic symptoms |
| XaCHs | All | [X] Single episode major depression without psychotic symptoms |
| XaCIs | All | Mild depression |
| XaCIt | All | Moderate depression |
| XaCIu | All | Severe depression |
| SNOMED Code | Term ID | Description |
| 832007' | | Moderate major depression (disorder) |
| 2618002' | | Chronic recurrent major depressive disorder (disorder) |
| 14070001' | | Multi-infarct dementia with depression (disorder) |
| 1.44.000.001 | | |
| 14183003' | | Chronic major depressive disorder, single episode (disorder) |
| 14183003 | | Chronic major depressive disorder, single episode (disorder) Severe recurrent major depression with psychotic features, mood-incongruent |
| 15193003' | | |
| | | Severe recurrent major depression with psychotic features, mood-incongruent |
| 15193003' | | Severe recurrent major depression with psychotic features, mood-incongruent (disorder) |
| 15193003'<br>15639000' | | Severe recurrent major depression with psychotic features, mood-incongruent (disorder) Moderate major depression, single episode (disorder) |
| 15193003'<br>15639000'<br>18818009'<br>19527009' | | Severe recurrent major depression with psychotic features, mood-incongruent (disorder) Moderate major depression, single episode (disorder) Moderate recurrent major depression (disorder) Single episode of major depression in full remission (disorder) Severe major depression, single episode, with psychotic features, mood- |
| 15193003'<br>15639000'<br>18818009' | | Severe recurrent major depression with psychotic features, mood-incongruent (disorder) Moderate major depression, single episode (disorder) Moderate recurrent major depression (disorder) Single episode of major depression in full remission (disorder) |
| 15193003'<br>15639000'<br>18818009'<br>19527009' | | Severe recurrent major depression with psychotic features, mood-incongruent (disorder) Moderate major depression, single episode (disorder) Moderate recurrent major depression (disorder) Single episode of major depression in full remission (disorder) Severe major depression, single episode, with psychotic features, mood- |

| 30605009' | Major depression in partial remission (disorder) |
|---|---|
| | Severe recurrent major depression with psychotic features, mood-congruent |
| 33078009' | (disorder) |
| 33135002' | Recurrent major depression in partial remission (disorder) |
| 33736005' | Severe major depression with psychotic features, mood-congruent (disorder) |
| 35489007' | Depressive disorder (disorder) |
| 36474008' | Severe recurrent major depression without psychotic features (disorder) |
| 36923009' | Major depression, single episode (disorder) |
| 38694004' | Recurrent major depressive disorder with atypical features (disorder) |
| 39809009' | Recurrent major depressive disorder with catatonic features (disorder) |
| 40379007' | Mild recurrent major depression (disorder) |
| 40568001' | Recurrent brief depressive disorder (disorder) |
| 42925002' | Major depressive disorder, single episode with atypical features (disorder) |
| 48589009' | Minor depressive disorder (disorder) |
| 58703003' | Postpartum depression (disorder) |
| 60099002' | Severe major depression with psychotic features, mood-incongruent (disorder) |
| 66344007' | Recurrent major depression (disorder) |
| 69392006' | Major depressive disorder, single episode with catatonic features (disorder) |
| 70747007' | Major depression single episode, in partial remission (disorder) |
| 71336009' | Recurrent major depressive disorder with postpartum onset (disorder) |
| 73867007' | Severe major depression with psychotic features (disorder) |
| 75084000' | Severe major depression without psychotic features (disorder) |
| 76441001' | Severe major depression, single episode, without psychotic features (disorder) |
| | Severe major depression, single episode, with psychotic features, mood- |
| 77911002' | congruent (disorder) |
| 79298009' | Mild major depression, single episode (disorder) |
| 79842004' | Stuporous depression (disorder) |

| 82218004' | Postoperative depression (disorder) |
|---|---|
| 83458005' | Agitated depression (disorder) |
| 87414006' | Reactive depression (situational) (disorder) |
| 87512008' | Mild major depression (disorder) |
| 161469008' | History of depression (situation) |
| 191495003' | Drug-induced depressive state (disorder) |
| 191604000' | Single major depressive episode, severe, with psychosis (disorder) |
| 191610000' | Recurrent major depressive episodes, mild (disorder) |
| 191611001' | Recurrent major depressive episodes, moderate (disorder) |
| 191613003' | Recurrent major depressive episodes, severe, with psychosis (disorder) |
| 191616006' | Recurrent depression (disorder) |
| 191659001' | Atypical depressive disorder (disorder) |
| 191676002' | Reactive depressive psychosis (disorder) |
| 192046006' | Brief depressive adjustment reaction (disorder) |
| 192049004' | Prolonged depressive adjustment reaction (disorder) |
| 192079006' | Postviral depression (disorder) |
| 192080009' | Chronic depression (disorder) |
| 231485007' | Post-schizophrenic depression (disorder) |
| 231499006' | Endogenous depression first episode (disorder) |
| 231500002' | Masked depression (disorder) |
| 231504006' | Mixed anxiety and depressive disorder (disorder) |
| 237349002' | Mild postnatal depression (disorder) |
| 237350002' | Severe postnatal depression (disorder) |
| 237739002' | Pseudo-Cushing's syndrome of depression (disorder) |
| 247803002' | Seasonal affective disorder (disorder) |
| 268621008' | Recurrent major depressive episodes (disorder) |

| 272022009' | Complaining of feeling depressed (finding) |
|---|---|
| 274948002' | Endogenous depression - recurrent (disorder) |
| 300706003' | Endogenous depression (disorder) |
| 310495003' | Mild depression (disorder) |
| 310496002' | Moderate depression (disorder) |
| 310497006' | Severe depression (disorder) |
| 319768000' | Recurrent major depressive disorder with melancholic features (disorder) |
| 320751009' | Major depression, melancholic type (disorder) |
| 321717001' | Involutional depression (disorder) |
| 366979004' | Depressed mood (finding) |
| 370143000' | Major depressive disorder (disorder) |
| 394924000' | Symptoms of depression (finding) |
| 395072006' | Counseling for postnatal depression (procedure) |
| 430852001' | Severe major depression, single episode, with psychotic features (disorder) |
| 450714000' | Severe major depression (disorder) |
| 704678007' | Depressed mood with postpartum onset (finding) |
| 712823008' | Acute depression (disorder) |
| 718636001' | Minimal depression (disorder) |
| 719592004' | Moderately severe major depression (disorder) |
| 719593009' | Moderately severe depression (disorder) |
| 720451004' | Minimal recurrent major depression (disorder) |
| 720452006' | Moderately severe recurrent major depression (disorder) |
| 720453001' | Moderately severe major depression single episode (disorder) |
| 720454007' | Minimal major depression single episode (disorder) |
| 720455008' | Minimal major depression (disorder) |
| 723928009' | Mood disorder with depressive symptoms caused by alcohol (disorder) |

| | Mood disorder with mixed manic and depressive symptoms caused by alcohol |
|---|---|
| 723930006' | (disorder) |
| 724676000' | Mood disorder with depressive symptoms caused by sedative (disorder) |
| 724677009' | Mood disorder with depressive symptoms caused by hypnotic (disorder) |
| 724678004' | Mood disorder with depressive symptoms caused by anxiolytic (disorder) |
| 724690002' | Mood disorder with depressive symptoms caused by cocaine (disorder) |
| 724757005' | Depressive symptoms due to primary psychotic disorder (disorder) |
| 726772006' | Major depression with psychotic features (disorder) |
| 762321000' | Mood disorder with depressive symptoms caused by opioid (disorder) |
| 762329003' | Mood disorder with depressive symptoms caused by stimulant (disorder) |
| 762336002' | Mood disorder with depressive symptoms caused by hallucinogen (disorder) |
| 762339009' | Mood disorder with depressive symptoms caused by volatile inhalant (disorder) |
| | Mood disorder with depressive symptoms caused by synthetic cathinone |
| 762512002' | (disorder) |
| 768835002' | Depression care management (procedure) |
| 788120007' | Antenatal depression (disorder) |
| | Mood disorder with mixed depressive and manic symptoms caused by |
| 838529004' | amfetamine and amfetamine derivative (disorder) |
| 871840004' | Episode of depression (finding) |
| 251000119105' | Severe major depression, single episode (disorder) |
| 281000119103' | Severe recurrent major depression (disorder) |
| 10211000132109' | Perinatal depression (disorder) |
| 94631000119100' | Depressive disorder in mother complicating pregnancy (disorder) |
| 133121000119109' | Severe seasonal affective disorder (disorder) |
| 199111000000100' | Referral for guided self-help for depression (procedure) |
| 286711000000107' | Counseling for depression (procedure) |
| 288751000119101' | Reactive depressive psychosis, single episode (disorder) |

| 361761000000106' | On full dose long term treatment for depression (finding) |
|---|---|
| 755321000000106' | Single major depressive episode, severe, with psychosis, psychosis in remission (disorder) |
| | Recurrent major depressive episodes, severe, with psychosis, psychosis in |
| 755331000000108' | remission (disorder) |
| 764611000000100' | Recurrent major depressive episodes, severe (disorder) |
| 764691000000109' | Recurrent major depressive episodes, in partial remission (disorder) |
| 764701000000109' | Recurrent major depressive episodes, in remission (disorder) |
| 764711000000106' | Single major depressive episode, in remission (disorder) |
| 923921000000104' | Referral for depression self-help video (procedure) |
| 1086471000000100' | Recurrent reactive depressive episodes, severe, with psychosis (disorder) |
| 1086661000000100' | Reactive depression, prolonged single episode (disorder) |
| 1086671000000100' | Reactive depression, single episode (disorder) |
| 1086681000000100' | Reactive depression, recurrent (disorder) |
| 1086691000000100' | Reactive depression, first episode (disorder) |
| 1089511000000100' | Recurrent depression with current severe episode and psychotic features (disorder) |
| 1089631000000100' | Recurrent depression with current severe episode without psychotic features (disorder) |
| 1089641000000100' | Recurrent depression with current moderate episode (disorder) |
| 10811121000119100' | Major depressive disorder in mother complicating childbirth (disorder) |
| 10811161000119100' | Major depressive disorder in mother complicating pregnancy (disorder) |
| 10835871000119100' | Depressive disorder in mother complicating childbirth (disorder) |
| 16238181000119100' | Depressive disorder caused by amphetamine (disorder) |
| 16238221000119100' | Depressive disorder caused by methamphetamine (disorder) |
| 16264621000119100' | Recurrent mild major depressive disorder co-occurrent with anxiety (disorder) |
| 16264821000119100' | Recurrent severe major depressive disorder co-occurrent with anxiety (disorder) |

| | | Recurrent moderate major depressive disorder co-occurrent with anxiety |
|---|---|---|
| 16264901000119100' | | (disorder) |
| 16265301000119100' | | Recurrent major depressive disorder in partial remission co-occurrent with anxiety (disorder) |
| 16265951000119100' | | Mild major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266831000119100' | | Moderate major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266991000119100' | | Severe major depressive disorder co-occurrent with anxiety single episode (disorder) |
| Recurrent depressive disorder | | |
| Read V2 Code | Term ID | Description |
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E2B1. | All | Chronic depression |
| | | [X]Recurrent major depressive episodes, severe, with psychosis, psychosis in |
| Eu32A | All | remission |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |

| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
|---|---|---|
| | | [X]Recurrent depressive disorder, current episode severe without psychotic |
| Eu332 | All | symptoms |
| | | [X]Recurrent depressive disorder, current episode severe with psychotic |
| Eu333 | All | symptoms |
| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Read CTV3 Code | Term ID | Description |
| Xa0wV | All | Recurrent brief depressive disorder |
| XM1GC | All | Endogenous depression - recurrent |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| | | Recurrent major depressive episodes, severe, with psychosis, psychosis in |
| XaX54 | All | remission |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |
| E1137 | All | Recurrent depression |
| E2B1. | All | Chronic depression |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| XE1Y1 | All | Recurrent major depressive episodes |
| | | [X]Recurrent depressive disorder, current episode severe without psychotic |
| XE1Zd | All | symptoms |

| | | [X]Recurrent depressive disorder, current episode severe with psychotic |
|---|---|---|
| XE1Ze | All | symptoms |
| XE1Zf | All | [X]Recurrent depressive disorder, unspecified |
| SNOMED Code | Term ID | Description |
| 15193003' | | Severe recurrent major depression with psychotic features, mood-incongruent (disorder) |
| 16264621000119100' | | Recurrent mild major depressive disorder co-occurrent with anxiety (disorder) |
| 16264821000119100' | | Recurrent severe major depressive disorder co-occurrent with anxiety (disorder) |
| 16264901000119100' | | Recurrent moderate major depressive disorder co-occurrent with anxiety (disorder) |
| 16265061000119100' | | Recurrent major depressive disorder co-occurrent with anxiety in full remission (disorder) |
| 16265301000119100' | | Recurrent major depressive disorder in partial remission co-occurrent with anxiety (disorder) |
| 18818009' | | Moderate recurrent major depression (disorder) |
| 191610000' | | Recurrent major depressive episodes, mild (disorder) |
| 191611001' | | Recurrent major depressive episodes, moderate (disorder) |
| 191613003' | | Recurrent major depressive episodes, severe, with psychosis (disorder) |
| 2618002' | | Chronic recurrent major depressive disorder (disorder) |
| 268621008' | | Recurrent major depressive episodes (disorder) |
| 274948002' | | Endogenous depression - recurrent (disorder) |
| 281000119103' | | Severe recurrent major depression (disorder) |
| 28475009' | | Severe recurrent major depression with psychotic features (disorder) |
| 319768000' | | Recurrent major depressive disorder with melancholic features (disorder) |
| 33078009' | | Severe recurrent major depression with psychotic features, mood-congruent (disorder) |
| 33135002' | | Recurrent major depression in partial remission (disorder) |

| 36474008' | | Severe recurrent major depression without psychotic features (disorder) |
|---|---|---|
| 38694004' | | Recurrent major depressive disorder with atypical features (disorder) |
| 39809009' | | Recurrent major depressive disorder with catatonic features (disorder) |
| 40379007' | | Mild recurrent major depression (disorder) |
| 66344007' | | Recurrent major depression (disorder) |
| 68019004' | | Recurrent major depression in remission (disorder) |
| 71336009' | | Recurrent major depressive disorder with postpartum onset (disorder) |
| 720451004' | | Minimal recurrent major depression (disorder) |
| 720452006' | | Moderately severe recurrent major depression (disorder) |
| | | Recurrent major depressive episodes, severe, with psychosis, psychosis in |
| 755331000000108' | | remission (disorder) |
| 764611000000100' | | Recurrent major depressive episodes, severe (disorder) |
| 764691000000109' | | Recurrent major depressive episodes, in partial remission (disorder) |
| 764701000000109' | | Recurrent major depressive episodes, in remission (disorder) |
| Depressive symptoms | | |
| Read V2 Code | Term ID | Description |
| 1B17. | All | Depressed |
| 1B1U. | All | Symptoms of depression |
| 1BQ | All | Loss of capacity for enjoyment |
| 1BT | All | Depressed mood |
| 1BU | All | Loss of hope for the future |
| 2257 | All | O/E - depressed |
| Read CTV3 Code | Term ID | Description |
| XE0re | All | Depressed mood |
| XaImU | All | Symptoms of depression |
| X761E | All | Loss of capacity for enjoyment |

| X761G | All | Loss of hope for the future |
|-------------------|---------|-----------------------------------------------|
| Xa3Xh | All | Feeling of hopelessness |
| 2257.' | All | O/E - depressed |
| XM0CR | All | C/O - feeling depressed |
| X00SO | All | Depressed |
| XaAyM | All | Feeling hopeless |
| SNOMED Code | Term ID | Description |
| 162722001' | | On examination - depressed (disorder) |
| 366979004' | | Depressed mood (finding) |
| 272022009' | | Complaining of feeling depressed (finding) |
| 307077003' | | Feeling hopeless (finding) |
| 1074741000000100' | | Unable to be hopeful for future (finding) |
| 1069851000000100' | | Difficulty being hopeful for future (finding) |
| 28669007' | | Anhedonia (finding) |
| 309838005' | | Emotional upset (finding) |
| 225014007' | | Feeling empty (finding) |
| 225457007' | | Feeling suicidal (finding) |
| 247796005' | | Loss of capacity for enjoyment (finding) |
| 430641005' | | Markedly diminished pleasure (finding) |
| 310480000' | | Complaining of tearfulness (finding) |
| 17029006' | | Feeling despair (finding) |
| 735640004' | | Excessive crying of adult (finding) |
| 271951008' | | Crying associated with mood (finding) |
| 394924000' | | Symptoms of depression (finding) |
| Parasuicide | | |
| Read V2 Code | Term ID | Description |

| U21 | All | [X]Intent self harm by hanging, strangulation/suffocation |
|---|---|---|
| U210. | All | [X]Int self harm by hanging, strangulation/suffocation occ home |
| U211. | All | [X]Intent self harm by hanging, strangulation/suffocation at res institut |
| U212. | All | [X]Int self harm by hanging, strangulation/suffocation in school/pub admin area |
| U213. | All | [X]Intent self harm by hanging, strangulation/suffocation in sport/athletic area |
| U214. | All | [X]Int self harm by hanging, strangulation/suffocation in street/highway |
| U215. | All | [X]Intent self harm by hanging, strangulation/suffocation trade/service area |
| U216. | All | [X]Int self harm by hanging, strangulation/suffocation indust/construct area |
| U217. | All | [X]Int self harm by hanging, strangulation/suffocation occ farm |
| U21y. | All | [X]Int self harm by hanging, strangulation/suffocation other spec place |
| U21z. | All | [X]Intent self harm by hanging, strangulation/suffocation unspecif place |
| U22 | All | [X]Intent self harm by drowning and submersion |
| U220. | All | [X]Int self harm by drowning and submersion occ home |
| U221. | All | [X]Intent self harm by drowning and submersion at res institut |
| U222. | All | [X]Int self harm by drowning and submersion in school/pub admin area |
| U223. | All | [X]Intent self harm by drowning and submersion in sport/athletic area |
| U224. | All | [X]Int self harm by drowning and submersion in street/highway |
| U225. | All | [X]Intent self harm by drowning and submersion trade/service area |
| U226. | All | [X]Int self harm by drowning and submersion indust/construct area |
| U227. | All | [X]Int self harm by drowning and submersion occ farm |
| U22y. | All | [X]Int self harm by drowning and submersion other spec place |
| U22z. | All | [X]Intent self harm by drowning and submersion unspecif place |
| U23 | All | [X]Intent self harm by handgun discharge |
| U230. | All | [X]Int self harm by handgun discharge occ home |
| U231. | All | [X]Intent self harm by handgun discharge at res institut |
| U232. | All | [X]Int self harm by handgun discharge in school/pub admin area |

| U233. | All | [X]Intent self harm by handgun discharge in sport/athletic area |
|---|---|---|
| U234. | All | [X]Int self harm by handgun discharge in street/highway |
| U235. | All | [X]Intent self harm by handgun discharge trade/service area |
| U236. | All | [X]Int self harm by handgun discharge indust/construct area |
| U237. | All | [X]Int self harm by handgun discharge occ farm |
| U23y. | All | [X]Int self harm by handgun discharge other spec place |
| U23z. | All | [X]Intent self harm by handgun discharge unspecif place |
| U24 | All | [X]Intentional self harm by rifle, shotgun and larger firearm discharge |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U240. | All | at home |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U241. | All | in residential institution |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U242. | All | at school, other institution and public administrative area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U243. | All | at sports and athletics area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U244. | All | on street and highway |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U245. | All | at trade and service area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U246. | All | at industrial and construction area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U247. | All | on farm |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U24y. | All | at other specified place |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U24z. | All | at unspecified place |

| U25 | All | [X]Intentional self harm by other and unspecified firearm discharge |
|---|---|---|
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U250. | All | at home |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U251. | All | in residential institution |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U252. | All | at school, other institution and public administrative area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U253. | All | at sports and athletics area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U254. | All | on street and highway |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U255. | All | at trade and service area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U256. | All | at industrial and construction area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U257. | All | on farm |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U25y. | All | at other specified place |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U25z. | All | at unspecified place |
| 2 | All | [X]Suicide |
| TK | All | Attempted suicide |
| TK0 | All | Suicide and selfinflicted poisoning by solid and liquid substances |
| TK00. | All | Suicide and selfinflicted poisoning by analgesics, antipyretics and anti-rheumatics |
| TK01. | All | Suicide + selfinflicted poisoning by barbiturates |
| TK010 | All | Suicide and self inflicted injury by Amylobarbitone |
| TK011 | All | Suicide and self inflicted injury by Barbitone |

| TK012 | All | Suicide and self inflicted injury by Butabarbitone |
|---|---|---|
| TK013 | All | Suicide and self inflicted injury by Pentabarbitone |
| TK014 | All | Suicide and self inflicted injury by Phenobarbitone |
| TK015 | All | Suicide and self inflicted injury by Quinalbarbitone |
| TK01z | All | Suicide and self inflicted injury by barbiturates |
| TK02. | All | Suicide and selfinflicted poisoning by other sedatives and hypnotics |
| TK03. | All | Suicide and selfinflicted poisoning by tranquillisers and other psychotropic |
| TK04. | All | agents Cylinde and colfinflicted poisoning by other drugg and medicines |
| | | Suicide and selfinflicted poisoning by other drugs and medicines |
| TK05. | All | Suicide + selfinflicted poisoning by drug or medicine NOS |
| my o c | A 11 | Suicide and selfinflicted poisoning by agricultural and horticultural chemical and |
| TK06. | All | pharmaceutical preparations other than plant foods and fertilizers |
| TK07. | All | Suicide and selfinflicted poisoning by corrosive and caustic substances |
| TK08. | All | Suicide and selfinflicted poisoning by arsenic and its compounds |
| TK0z. | All | Suicide and selfinflicted poisoning by solid and liquid substances NOS |
| TK1 | All | Suicide + selfinflicted poisoning by gases in domestic use |
| TK10. | All | Suicide and selfinflicted poisoning by gas distributed by pipeline |
| | | Suicide and selfinflicted poisoning by liquefied petroleum gas distributed in |
| TK11. | All | mobile containers |
| TK1y. | All | Suicide and selfinflicted poisoning by other utility gas |
| TK1z. | All | Suicide and selfinflicted poisoning by gases in domestic use NOS |
| TK2 | All | Suicide and selfinflicted poisoning by other gases and vapours |
| TK20. | All | Suicide and selfinflicted poisoning by motor vehicle exhaust gas |
| TK21. | All | Suicide and selfinflicted poisoning by other carbon monoxide |
| TK2y. | All | Suicide and selfinflicted poisoning by other gases and vapours |
| TK2z. | All | Suicide + selfinflicted poisoning by gases and vapours NOS |
| ТКЗ | All | Suicide and selfinflicted injury by hanging, strangulation and suffocation |

| TK31. | All | Suicide and selfinflicted injury by suffocation by plastic bag |
|---|---|---|
| | | Suicide and selfinflicted injury by other means of hanging, strangulation and |
| TK3y. | All | suffocation |
| TK3z. | All | Suicide and selfinflicted injury by hanging, strangulation and suffocation NOS |
| TK4 | All | Suicide and selfinflicted injury by drowning |
| TK5 | All | Suicide and selfinflicted injury by firearms and explosives |
| TK50. | All | Suicide and selfinflicted injury by handgun |
| TK51. | All | Suicide and selfinflicted injury by shotgun |
| TK52. | All | Suicide and selfinflicted injury by hunting rifle |
| TK53. | All | Suicide and selfinflicted injury by military firearms |
| TK54. | All | Suicide and selfinflicted injury by other firearm |
| TK55. | All | Suicide and selfinflicted injury by explosives |
| TK5z. | All | Suicide and selfinflicted injury by firearms and explosives NOS |
| TK6 | All | Suicide and selfinflicted injury by cutting and stabbing instruments |
| TK60. | All | Suicide and selfinflicted injury by cutting |
| TK61. | All | Suicide and selfinflicted injury by stabbing |
| TK6z. | All | Suicide and selfinflicted injury by cutting and stabbing instruments NOS |
| TK7 | All | Suicide and selfinflicted injury by jumping from high place |
| TK70. | All | Suicide and selfinflicted injury by jumping from residential premises |
| TK71. | All | Suicide and selfinflicted injury by jumping from other manmade structure |
| TK72. | All | Suicide and selfinflicted injury by jumping from natural sites |
| TK72. | All | Suicide and selfinflicted injury by jumping from natural sites |
| TK7z. | All | Suicide and selfinflicted injury by jumping from high place NOS |
| TKx | All | Suicide and selfinflicted injury by other means |
| TKx0. | All | Suicide and selfinflicted injury by jumping or lying before moving object |
| TKx01 | All | Suicide and selfinflicted injury by lying before moving object |

| TKx0z | All | Suicide and selfinflicted injury by jumping or lying before moving object NOS |
|---|---|---|
| TKx1. | All | Suicide and selfinflicted injury by burns or fire |
| TKx2. | All | Suicide and selfinflicted injury by scald |
| TKx3. | All | Suicide and selfinflicted injury by extremes of cold |
| TKx4. | All | Suicide and selfinflicted injury by electrocution |
| TKx5. | All | Suicide and selfinflicted injury by crashing of motor vehicle |
| TKx6. | All | Suicide and selfinflicted injury by crashing of aircraft |
| TKx7. | All | Suicide and selfinflicted injury by caustic substances, except poisoning |
| TKxy. | All | Suicide and selfinflicted injury by other specified means |
| TKxz. | All | Suicide and selfinflicted injury by other means NOS |
| TKz | All | Suicide and selfinflicted injury NOS |
| Read CTV3 Code | Term ID | Description |
| Xa04L | All | Parasuicide |
| Xa3jI | All | Attempted suicide NOS |
| 146A. | All | H/O: attempted suicide |
| XM1Fs | All | Self hanging, strangulation or suffocation |
| TK3 | All | Suicide and selfinflicted injury by hanging, strangulation and suffocation |
| TK30. | All | Suicide or attempted suicide by hanging |
| Xa3jC | All | Attempted suicide - hanging |
| Xa3jL | All | Suicide - hanging |
| | | Suicide and selfinflicted injury by other means of hanging, strangulation and |
| TK3y. | All | suffocation |
| TK3z. | All | Suicide and selfinflicted injury by hanging, strangulation and suffocation NOS |
| XE22I | All | Suicide and selfinflicted injury by suffocation by plastic bag |
| Xa3jD | All | Attempted suicide - suffocation |
| Xa3jM | All | Suicide - suffocation |

| TKO | All | Suicide and selfinflicted poisoning by solid and liquid substances |
|---|---|---|
| TK0z. | All | Suicide and selfinflicted poisoning by solid and liquid substances NOS |
| TK4 | All | Suicide and selfinflicted injury by drowning |
| TK5 | All | Suicide or selfinflicted injury by firearms and explosives |
| TK50. | All | Suicide or selfinflicted injury by handgun |
| TK51. | All | Suicide or selfinflicted injury by shotgun |
| TK52. | All | Suicide or selfinflicted injury by hunting rifle |
| TK53. | All | Suicide or selfinflicted injury by military firearm |
| TK54. | All | Suicide and selfinflicted injury by other firearm |
| TK55. | All | Suicide or selfinflicted injury by explosives |
| TK5z. | All | Suicide and selfinflicted injury by firearms and explosives NOS |
| Xa3jF | All | Attempted suicide - firearms |
| Xa3j0 | All | Suicide - firearms |
| TK6 | All | Suicide or selfinflicted injury by cutting and stabbing |
| TK60. | All | Suicide or selfinflicted injury by cutting |
| TK61. | All | Suicide or selfinflicted injury by stabbing |
| TK6z. | All | Suicide and selfinflicted injury by cutting and stabbing instruments NOS |
| Xa3jG | All | Attempted suicide - cut/stab |
| Xa3jP | All | Suicide - cut/stab |
| TK7 | All | Suicide or self injury by jumping from a height |
| TK70. | All | Suicide and selfinflicted injury by jumping from residential premises |
| TK71. | All | Suicide and selfinflicted injury by jumping from other man-made structure |
| TK72. | All | Suicide and selfinflicted injury by jumping from natural sites |
| TK72. | All | Suicide and selfinflicted injury by jumping from natural sites |
| TK7z. | All | Suicide and selfinflicted injury by jumping from high place NOS |
| X71B6 | All | Suicide or self injury by jumping from high man-made structure |
| VE4DE | 4.11 | |
|---|---|---|
| X71B7 | All | Suicide or self injury by jumping from high building |
| X71B8 | All | Suicide or self injury by jumping from bridge |
| X71B9 | All | Suicide or self injury by jumping from high natural feature |
| X71BA | All | Suicide or self injury by jumping off cliff |
| ХаЗјН | All | Attempted suicide - jumping from a high place |
| Xa3jQ | All | Suicide - jumping from a high place |
| TKx | All | Suicide and selfinflicted injury by other means |
| TKx0. | All | Suicide and selfinflicted injury by jumping or lying before moving object |
| TKx00 | All | Suicide and selfinflicted injury by jumping before moving object |
| TKx01 | All | Suicide and selfinflicted injury by lying before moving object |
| TKx0z | All | Suicide and selfinflicted injury by jumping or lying before moving object NOS |
| TKxy. | All | Suicide and selfinflicted injury by other specified means |
| TKxz. | All | Suicide and selfinflicted injury by other means NOS |
| TKx1. | All | Suicide or self injury by burning or fire |
| TKx2. | All | Suicide or self injury by scalding |
| X71BF | All | Suicide or self injury by igniting petrol soaked clothing |
| X71BG | All | Suicide or self injury by arson |
| TKx3. | All | Suicide or self injury by exposure to cold |
| TKx4. | All | Suicide or self injury by electric current |
| TKx7. | All | Suicide and selfinflicted injury by caustic substances, excluding poisoning |
| TKz | All | Suicide and selfinflicted injury NOS |
| Xa3jI | All | Attempted suicide NOS |
| Xa3jR | All | Suicide NOS |
| X71B3 | All | Self poisoning by gas |
| TK1 | All | Suicide and selfinflicted poisoning by gases in domestic use |
| TK21. | All | Suicide and selfinflicted poisoning by other carbon monoxide |

| TK2y. | All | Suicide and selfinflicted poisoning by other gases and vapours |
|---|---|---|
| TK2z. | All | Suicide and selfinflicted poisoning by gases and vapours NOS |
| X71B4 | All | Self poisoning by carbon monoxide |
| TK20. | All | Self poisoning by motor vehicle exhaust gas |
| X71B5 | All | Self poisoning by coal gas |
| X71BB | All | Suicide or self injury associated with moving vehicles |
| TKx5. | All | Suicide or selfinflicted injury by crashing motor vehicle |
| TKx6. | All | Suicide or selfinflicted injury by crashing of aircraft |
| X71BC | All | Suicide or self injury by placing self in path of moving vehicle |
| X71BD | All | Suicide or self injury by placing self in path of moving motor vehicle |
| X71BE | All | Suicide or self injury by placing self in path of moving railway vehicle |
| XE22J | All | Suicide or attempted suicide by drowning |
| Xa3jE | All | Attempted suicide - drowning |
| Xa3jN | All | Suicide - drowning |
| XM1Fs | All | Self hanging, strangulation or suffocation |
| TK3 | All | Suicide and selfinflicted injury by hanging, strangulation and suffocation |
| TK30. | All | Suicide or attempted suicide by hanging |
| Xa3jL | All | Suicide - hanging |
| | | Suicide and selfinflicted injury by other means of hanging, strangulation and |
| TK3y. | All | suffocation |
| TK3z. | All | Suicide and selfinflicted injury by hanging, strangulation and suffocation NOS |
| XE22I | All | Suicide and selfinflicted injury by suffocation by plastic bag |
| Xa3jD | All | Attempted suicide - suffocation |
| Xa3jM | All | Suicide - suffocation |
| TK50. | All | Suicide or selfinflicted injury by handgun |
| Ua1AA | All | Hanging self |

| Ua1AB | All | Drowning self |
|---|---|---|
| Ua1A9 | All | Jumping from height |
| Ua1A8 | All | Jumping from building |
| Ua1A7 | All | Jumping from bridge |
| Ua14U | All | Jumping from cliff |
| Ua1AE | All | Self-asphyxiation |
| Ua1AD | All | Self-strangulation |
| Ua1AC | All | Self-suffocation Self-suffocation |
| Ua14S | All | Throwing self in front of vehicle |
| Ua14T | All | Throwing self in front of train |
| X71B0 | All | Self poisoning by non-drug solid or liquid agents |
| TK07. | All | Self poisoning by corrosive or caustic substance |
| TK08. | All | Self poisoning by arsenic or its compounds |
| X71B2 | All | Self poisoning by plants or parts of plants |
| XM1FX | All | Self poisoning by agricultural chemical |
| | | Suicide and selfinflicted poisoning by agricultural and horticultural chemical and |
| TK06. | All | pharmaceutical preparations other than plant foods and fertilizers |
| X71B1 | All | Self poisoning by paraquat |
| Ua14R | All | Shooting self |
| Xa2pL | All | Stabbing self |
| U21 | All | [X]Intent self harm by hanging, strangulation/suffocation |
| U210. | All | [X]Int self harm by hanging, strangulation/suffocation occ home |
| U211. | All | [X]Intent self harm by hanging, strangulation/suffocation at res institut |
| U212. | All | [X]Int self harm by hanging, strangulation/suffocation in school/pub admin area |
| U213. | All | [X]Intent self harm by hanging, strangulation/suffocation in sport/athletic area |
| U214. | All | [X]Int self harm by hanging, strangulation/suffocation in street/highway |

| U215. | All | [X]Intent self harm by hanging, strangulation/suffocation trade/service area |
|---|---|---|
| U216. | All | [X]Int self harm by hanging, strangulation/suffocation indust/construct area |
| U217. | All | [X]Int self harm by hanging, strangulation/suffocation occ farm |
| U21y. | All | [X]Int self harm by hanging, strangulation/suffocation other spec place |
| U21z. | All | [X]Intent self harm by hanging, strangulation/suffocation unspecif place |
| U22 | All | [X]Intent self harm by drowning and submersion |
| U220. | All | [X]Int self harm by drowning and submersion occ home |
| U221. | All | [X]Intent self harm by drowning and submersion at res institut |
| U222. | All | [X]Int self harm by drowning and submersion in school/pub admin area |
| U223. | All | [X]Intent self harm by drowning and submersion in sport/athletic area |
| U224. | All | [X]Int self harm by drowning and submersion in street/highway |
| U225. | All | [X]Intent self harm by drowning and submersion trade/service area |
| U226. | All | [X]Int self harm by drowning and submersion indust/construct area |
| U227. | All | [X]Int self harm by drowning and submersion occ farm |
| U22y. | All | [X]Int self harm by drowning and submersion other spec place |
| U22z. | All | [X]Intent self harm by drowning and submersion unspecif place |
| U23 | All | [X]Intent self harm by handgun discharge |
| U230. | All | [X]Int self harm by handgun discharge occ home |
| U231. | All | [X]Intent self harm by handgun discharge at res institut |
| U232. | All | [X]Int self harm by handgun discharge in school/pub admin area |
| U233. | All | [X]Intent self harm by handgun discharge in sport/athletic area |
| U234. | All | [X]Int self harm by handgun discharge in street/highway |
| U235. | All | [X]Intent self harm by handgun discharge trade/service area |
| U236. | All | [X]Int self harm by handgun discharge indust/construct area |
| U237. | All | [X]Int self harm by handgun discharge occ farm |
| U23y. | All | [X]Int self harm by handgun discharge other spec place |

| U23z. | All | [X]Intent self harm by handgun discharge unspecif place |
|---|---|---|
| U24 | All | [X]Intentional self harm by rifle, shotgun and larger firearm discharge |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U240. | All | at home |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U241. | All | in residential institution |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U242. | All | at school, other institution and public administrative area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U243. | All | at sports and athletics area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U244. | All | on street and highway |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U245. | All | at trade and service area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U246. | All | at industrial and construction area |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U247. | All | on farm |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U24y. | All | at other specified place |
| | | [X]Intentional self harm by rifle, shotgun and larger firearm discharge, occurrence |
| U24z. | All | at unspecified place |
| U25 | All | [X]Intentional self harm by other and unspecified firearm discharge |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U250. | All | at home |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U251. | All | in residential institution |

| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
|---|---|---|
| U252. | All | at school, other institution and public administrative area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U253. | All | at sports and athletics area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U254. | All | on street and highway |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U255. | All | at trade and service area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U256. | All | at industrial and construction area |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U257. | All | on farm |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U25y. | All | at other specified place |
| | | [X]Intentional self harm by other and unspecified firearm discharge, occurrence |
| U25z. | All | at unspecified place |
| SNOMED Code | Term ID | Description |
| 225048008 | | Jumping from height (finding) |
| 225046007 | | Jumping from bridge (finding) |
| 225047003 | | Jumping from building (finding) |
| 224950008 | | Jumping from cliff (finding) |
| 224949008 | | Throwing self in front of train (finding) |
| 224948000 | | Throwing self in front of vehicle (finding) |
| 225049000 | | Hanging self (finding) |
| 428422006 | | Found hanging self (finding) |
| 161474000 | | History of attempted suicide (situation) |
| 82313006 | | Suicide attempt (event) |

| 269808005 | Attempt suicide - car exhaust (event) |
|---|---|
| 288311002 | Attempt suicide - domestic gas (event) |
| 287185009 | Attempted suicide - cut/stab (event) |
| 287183002 | Attempted suicide - drowning (event) |
| 287184008 | Attempted suicide - firearms (event) |
| 287181000 | Attempted suicide - hanging (event) |
| 287186005 | Attempted suicide - jumping from a high place (event) |
| 287182007 | Attempted suicide - suffocation (event) |
| 36153001 | First known suicide attempt (event) |
| 23233009 | Previous known suicide attempt (event) |
| 53846008 | Suicide attempt by adequate means (event) |
| 55554002 | Suicide attempt by inadequate means (event) |
| 219110007 | Suicide and self inflicted injury by amylobarbitone (navigational concept) |
| 269725004 | Suicide and selfinflicted injury (navigational concept) |
| 219141008 | Suicide and selfinflicted injury by drowning (navigational concept) |
| 219111006 | Suicide and self inflicted injury by Barbitone (navigational concept) |
| 219115002 | Suicide and self inflicted injury by Quinalbarbitone (navigational concept) |
| 219116001 | Suicide and self inflicted injury by barbiturates (navigational concept) |
| 219112004 | Suicide and self inflicted injury by Butabarbitone (navigational concept) |
| 219114003 | Suicide and self inflicted injury by phenobarbitone (navigational concept) |
| 219113009 | Suicide and self inflicted injury by Pentabarbitone (navigational concept) |
| 219150005 | Suicide or selfinflicted injury by cutting and stabbing (navigational concept) |
| 219142001 | Suicide or selfinflicted injury by firearms and explosives (navigational concept) |
| 219125007 | Suicide and selfinflicted poisoning by gases in domestic use (disorder) |
| 219126008 | Suicide and selfinflicted poisoning by gas distributed by pipeline (disorder) |

| | Suicide and selfinflicted poisoning by liquefied petroleum gas distributed in |
|---|---|
| 219127004 | mobile containers (disorder) |
| | Suicide and selfinflicted injury by suffocation by plastic bag (navigational |
| 269726003 | concept) |
| | Suicide and selfinflicted injury by jumping from natural sites (navigational |
| 219158003 | concept) |
| | Suicide and selfinflicted injury by lying before moving object (navigational |
| 219163004 | concept) |
| | Suicide and selfinflicted injury by jumping before moving object (navigational |
| 219162009 | concept) |
| | Suicide and selfinflicted injury by jumping from residential premises |
| 219156004 | (navigational concept) |
| | Suicide and selfinflicted injury by jumping or lying before moving object |
| 219161002 | (navigational concept) |
| | Suicide and selfinflicted injury by caustic substances, excluding poisoning |
| 219171000 | (navigational concept) |
| | Suicide and selfinflicted poisoning by analgesics, antipyretics and anti-rheumatics |
| 219108005 | (navigational concept) |
| 240407000 | Suicide and selfinflicted poisoning by solid and liquid substances (navigational |
| 219107000 | concept) |
| 240426000 | Suicide and selfinflicted injury by hanging, strangulation and suffocation |
| 219136000 | (navigational concept) |
| 27000002 | Patient suicide, or attempted suicide resulting in serious disability, while being |
| 370908002 | cared for in a healthcare facility (event) |
| 271982007 | Intentional self poisoning (disorder) |
| 363293009 | Self-administered poisoning (disorder) |
| 242839001 | Self poisoning by gas (disorder) |
| 242840004 | Self poisoning caused by carbon monoxide (disorder) |

| 242841000 | | Self poisoning caused by coal gas (disorder) |
|---|---|---|
| 219131005 | | Self poisoning caused by motor vehicle exhaust gas (disorder) |
| 242836008 | | Self poisoning by non-drug solid or liquid agents (disorder) |
| 274912004 | | Self poisoning by agricultural chemical (disorder) |
| 219122005 | | Self poisoning by corrosive or caustic substance (disorder) |
| 242837004 | | Self poisoning by paraquat (disorder) |
| 242838009 | | Self poisoning by plants or parts of plants (disorder) |
| 219123000 | | Self poisoning caused by arsenic or its compounds (disorder) |
| 284744004 | | Burning self (finding) |
| 307578000 | | Cutting own wrists (finding) |
| 225045006 | | Cutting own throat (finding) |
| 224947005 | | Shooting self (finding) |
| 284759005 | | Stabbing self (finding) |
| 219166007 | | Suicide or self injury by scalding (navigational concept) |
| 225050000 | | Drowning self (finding) |
| 219333004 | | Drowning or immersion of unknown intent (event) |
| 418765005 | | Exposure to potentially harmful entity, undetermined intent (event) |
| 219328003 | | Hanging, strangulation or suffocation of unknown intent (event) |
| 219329006 | | Hanging of unknown intent (event) |
| 219330001 | | Suffocation of unknown intent by plastic bag (event) |
| 219342006 | | Injury of unknown intent by sharp instrument (disorder) |
| Absence from school | | |
| Read V2 Code | Term ID | Description |
| E2C10 | All | School refusal |
| E2D2z | All | School refusal |
| 13Z4J | All | School attendance poor |

| Eu912 | All | [X]Truancy from school |
|---|---|---|
| E2C10 | All | Unsocial childhood truancy |
| E2C20 | All | Socialised childhood truancy |
| Read CTV3 Code | Term ID | Description |
| X766A | All | School refusal |
| 13Z4J | All | School attendance poor |
| X7667 | All | Intentional non-attendance at school |
| 13Z4G | All | Left school free will |
| X7669 | All | Parental withholding from school |
| X7668 | All | Truancy |
| XE1Yt | All | Unsocial childhood truancy |
| E2C20 | All | Socialised childhood truancy |
| SNOMED Code | Term ID | Description |
| 248050007 | | Intentional non-attendance at school (finding) |
| 248052004 | | School refusal (finding) |
| 105479008 | | Truancy (finding) |
| 248051006 | | Parental withholding from school (finding) |
| 161131005 | | Left school free will (finding) |
| 161133008 | | School attendance poor (finding) |
| 440680000 | | Unable to attend school due to illness (finding) |
| 31492004 | | Fear of school (finding) |
| 271947006 | | School phobia (finding) |
| Unemployment | | |
| Unemployment | | |
| Unemployment Read V2 Code | Term ID | Description |
| | Term ID | <b>Description</b> Unemployed |

| 13J71 | All | Chronic unemployment |
|---|---|---|
| ZV620 | All | [V]Unemployment |
| 13R | All | Unemployment benefits |
| 13R1. | All | Unemployment benefit |
| 13R2. | All | Redundancy payment |
| 13RZ. | All | Unemployment benefit NOS |
| 13JX. | All | Time off work |
| 13JG. | All | Voluntarily redundant |
| 13J3. | All | Loss of job |
| 13J30 | All | Sacked from work |
| 13J8. | All | Redundant |
| 13JJ. | All | Unfit for work |
| 13JJ0 | All | Benefit agency reports unfit for work |
| 13JJ1 | All | Benefit agency reports unfit for work but fit note no longer required |
| 13Jk. | All | Not in employment, education or training |
| 9DG4. | All | IB 113 DLS incapacity for work form paid |
| 9DG2. | All | IB 113 DLS incapacity for work form sent |
| 9DG3. | All | IB 113 DLS incapacity for work form received |
| 9DG1. | All | IB 113 DLS incapacity for work form completed |
| 9DQ3. | All | ESA113 form paid |
| 9DQ1. | All | ESA113 form sent |
| 9DQ2. | All | ESA113 form received |
| 9DQ0. | All | ESA113 form completed |
| 130D. | All | Employment and support allowance |
| Read CTV3 Code | Term ID | Description |
| 13J7. | All | Unemployed |

| 13J70 | All | Recently unemployed |
|---|---|---|
| 13J71 | All | Chronic unemployment |
| ZV620 | All | [V]Unemployment |
| XaPhf | All | Benefit agency reports unfit for work |
| Xabd4 | All | Benefit agency reports unfit for work but fit note no longer required |
| 13J8. | All | Redundant |
| 13JG. | All | Voluntarily redundant |
| Ua2BD | All | Unfit to return to work |
| Ua2BE | All | Physically unfit for work |
| U12BF | All | Mentally unfit for work |
| 13JX. | All | Time off work |
| XaZHu | All | ESA113 form paid |
| XaZHt | All | ESA113 form sent |
| XaZHs | All | ESA113 form received |
| XaZHj | All | ESA113 form completed |
| XaBhC | All | Employment and support allowance |
| XacJr | All | Not in employment, education or training |
| XE0pT | All | Loss of job |
| Ua0V9 | All | Dismissed from job |
| Ua0VA | All | Unfair dismissal from job |
| XaClW | All | IB 113 DLS incapacity for work form paid |
| XaCIU | All | IB 113 DLS incapacity for work form sent |
| XaCIV | All | IB 113 DLS incapacity for work form received |
| XaCIT | All | IB 113 DLS incapacity for work form completed |
| 13JJ. | All | Unfit for work |
| 13J6. | All | Medically retired |

| SNOMED Code | Term ID | Description |
|---|---|---|
| 266956001 | | Loss of job (finding) |
| 105496009 | | Dismissed from job (finding) |
| 160901009 | | Made redundant (finding) |
| 73438004 | | Unemployed (finding) |
| 160900005 | | Chronic unemployment (finding) |
| 160899000 | | Recently unemployed (finding) |
| 354581000000101' | | Unemployed person (person) |
| 719401000000102' | | Unemployed person (qualifier value) |
| 224474004 | | Unfair dismissal from job (finding) |
| 105498005 | | Voluntarily redundant (finding) |
| 723481000000104' | | Youth unemployment (qualifier value) |
| 161005005 | | Unemployment benefits (qualifier value) |
| 161006006 | | Unemployment benefit (qualifier value) |
| 723971000000106' | | Long term unemployment (qualifier value) |
| 313083007 | | Unemployment counseling (procedure) |
| 313084001 | | Redundancy counseling (procedure) |
| 281559009 | | Number of days off work (observable entity) |
| 160928004 | | Amount of time off work (observable entity) |
| 439907006 | | Number of sick days off work in last month (observable entity) |
| 105495008 | | Forced retirement, life event (finding) |
| 925481000000108' | | Benefits agency reports unfit for work but fit note no longer needed (finding) |
| 161007002 | | Redundancy payment (qualifier value) |
| 160910001 | | Unfit for work (finding) |
| 374171000000109' | | Benefits agency reports unfit for work (finding) |
| 304248001 | | Unfit for particular post (finding) |

| 225888002 | | Unfit to return to work (finding) |
|---|---|---|
| 225890001 | | Mentally unfit to return to work (finding) |
| 225889005 | | Physically unfit to return to work (finding) |
| 224384002 | | Registered with job center (finding) |
| 224385001 | | Registered with work placement officer (finding) |
| 14121000000104' | | IB113 DLS Incapacity for work form sent (finding) |
| 14141000000106' | | IB113 DLS Incapacity for work form paid (finding) |
| 14131000000102' | | IB113 DLS Incapacity for work form received (finding) |
| 14111000000105' | | IB113 DLS Incapacity for work form completed (finding) |
| 835611000000109' | | Employment and support allowance status (finding) |
| 835641000000105' | | Employment and support allowance 113 form completed (finding) |
| 835711000000103' | | Employment and support allowance 113 form paid (finding) |
| 835691000000100' | | Employment and support allowance 113 form received (finding) |
| 835671000000104' | | Employment and support allowance 113 form sent (finding) |
| 957481000000103' | | Not in employment, education or training (finding) |
| Absence from work | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| IBD symptoms - abdominal pain | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| IBD symptoms - discomforts or bloating | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |

| SNOMED Code | Term ID | Description |
|----------------------------------|---------|-------------|
| IBD symptoms - diarrhoea | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| IBD symptoms - weight loss | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| IBD symptoms - tiredness/fatigue | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Growth retardation related codes | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |

**sTable 3.2** Read and SNOMED codes to be used to identify the severity of IBD

| Medication use | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Surgical intervention | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Hospital admissions | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |
| Nutritional supplements (Modulen, Fortisip, Ensure, Osmolite, and Neocate) | | |
| Read V2 Code | Term ID | Description |
| Read CTV3 Code | Term ID | Description |
| SNOMED Code | Term ID | Description |